# Foundation Fighting Blindness (FFB) Consortium

<u>Universal Rare</u> Gene Study: A Registry and Natural History Study of Retinal Dystrophies Associated with Rare Disease-Causing Genetic Variants

**Protocol Identifying Number:** Uni-Rare **Funded by:** Foundation Fighting Blindness

Version Number: 1.2 12DEC2022

## **Key Roles and Signature Page**<u>Uni</u>versal <u>Rare</u> Gene Study

Protocol Identifying Number: Uni-Rare

Version Number: v1.2 12DEC2022

| Protocol Chair | |
|-----------------------------|-----------------------------|
| Name, degree | José-Alain Sahel, M.D. |
| Signature/Date | |
| JCHR Protocol Director (Spo | onsor) |
| Name, degree | Allison Ayala, MS |
| Signature/Date | |
| FFB Representative (Funder) | |
| Name, degree | Todd Durham, PhD. |
| Signature/Date | |
| Statistician | |
| Name, degree | Maureen Maguire, PhD, FARVO |
| Signature/Date | |

## TABLE OF CONTENTS

| CHAPTER 1: BACKGROUND INFORMATION | 23 |
|------------------------------------------------------------------------|----|
| 1.1 Introduction | 23 |
| 1.1.1 Identifying Optimal IRD Patient Populations for Target Therapies | 23 |
| 1.1.2 Develop and Validate Outcome Measures for Progression of IRDs | 23 |
| 1.1.3 Other Gaps Addressed by Natural History Studies | 24 |
| 1.1.4 Unique Challenges in Ultra-Rare Genes | 24 |
| 1.2 Rationale for a Universal Rare Gene Study | 24 |
| 1.3 Study Objectives | 25 |
| 1.4 Potential Risks and Benefits | 26 |
| 1.4.1 Known Potential Risks | 26 |
| 1.4.2 Known Potential Benefits | 26 |
| 1.4.3 Risk Assessment | 27 |
| 1.5 General Considerations | 27 |
| CHAPTER 2: REGISTRY ENROLLMENT AND REGISTRY/SCREENING VISIT | |
| 2.1 Registry Recruitment and Enrollment | |
| 2.2 Cohort Definitions | 28 |
| 2.3 Registry Informed Consent and Authorization Procedures | 29 |
| 2.4 Registry/Screening Visit | 31 |
| 2.4.1 Registry Eligibility Criteria | 31 |
| 2.4.1.1 Participant Inclusion Criteria | 31 |
| 2.4.1.2 Ocular Inclusion Criteria | 32 |
| 2.4.1.3 Participant Exclusion Criteria | 32 |
| 2.4.1.4 Ocular Exclusion Criteria | 32 |
| 2.4.2 Registry/Screening Visit Data Collection and Testing | 33 |
| 2.4.3 Initial Screen Failures | |
| 2.5 Genetic Screening Phase | 35 |
| 2.5.1 Genetic Screen Failures | 35 |
| 2.5.2 Genetics Committee Review | 36 |
| 2.6 Final Registry Cohort Criteria | 36 |
| CHAPTER 3: REGISTRY PHASE | 37 |
| 3.1 Evaluation of Natural History Study (NHS) Target Gene Status | 37 |
| 3.2 Annual Phone Calls | 37 |
| 3.3 Completion of Registry Phase | 37 |
| CHAPTER 4: NATURAL HISTORY STUDY ENROLLMENT AND BASELINE VISIT | 38 |

| 4.1 Natural History Study (NHS) Target Gene Selection | 38 |
|--------------------------------------------------------------|----|
| 4.2 NHS Enrollment | 38 |
| 4.2.1 NHS Informed Consent and Authorization Procedures | 38 |
| 4.2.2 NHS Eligibility Criteria | 39 |
| 4.3 Baseline Visit Testing Procedures | 39 |
| 4.3.1 Younger Age Cohort | 40 |
| 4.3.2 Vision Cohorts 1 & 2 | 41 |
| 4.3.3 Vision Cohort 3 | 43 |
| CHAPTER 5: NATURAL HISTORY STUDY FOLLOW-UP VISITS | |
| 5.1 Follow-up Schedule | |
| 5.2 Target Timelines | |
| 5.3 Follow-up Visit Testing Procedures | |
| 5.3.1 Younger Age Cohort | |
| 5.3.1.1 Age-Up Procedures | |
| 5.3.2 Vision Cohorts 1 & 2 | |
| 5.3.3 Vision Cohort 3 | 48 |
| 5.3.4 Unscheduled Visits | 49 |
| CHAPTER 6: TESTING PROCEDURES AND QUESTIONNAIRES | |
| 6.1 Study Procedure Requirements | |
| 6.2 Questionnaires | 52 |
| CHAPTER 7: UNANTICIPATED PROBLEM AND ADVERSE EVENT REPORTING | 54 |
| 7.1 Unanticipated Problems | 54 |
| 7.2 Adverse Events | 54 |
| 7.2.1 Definitions | 54 |
| 7.2.2 Reportable Adverse Events | 55 |
| 7.2.3 Relationship of Adverse Event to Study Procedure | |
| 7.2.4 Severity (Intensity) of Adverse Event | |
| 7.2.5 Expectedness | |
| 7.2.6 Coding of Adverse Events | |
| 7.2.7 Outcome of Adverse Event | |
| 7.3 Timing of Event Reporting | 57 |
| CHAPTER 8: MISCELLANEOUS CONSIDERATIONS | |
| 8.1 New or Ongoing Medical Conditions and Medications | |
| 8.1.1 Pre-Existing Conditions | |
| 9.1.2 Madigations | 50 |

| 8.1.3 Medical Conditions During the Natural History Study | 58 |
|---|---|
| 8.2 Prohibited Medications, Treatments, and Procedures During the Natural History Study | 58 |
| 8.2.1 Prohibited Medications and Treatment for Retinal Degeneration | 58 |
| 8.2.2 Intraocular Surgical Procedures | 58 |
| 8.2.3 Treatment for Cystoid Macular Edema (CME) | 59 |
| 8.3 Pregnancy Reporting | 59 |
| 8.4 Participant Compensation | 59 |
| 8.5 Participant Withdrawal | 59 |
| 8.6 Confidentiality | 59 |
| CHAPTER 9: STATISTICAL CONSIDERATIONS | 60 |
| 9.1 Sample Size Approach | 60 |
| 9.1.1 General Considerations | 60 |
| 9.1.2 Registry Sample Size Considerations | 60 |
| 9.1.3 Natural History Study Sample Size Considerations | 62 |
| 9.2 Data Analysis | 67 |
| 9.2.1 Registry Data Analysis | 67 |
| 9.2.2 Natural History Data Analysis | 68 |
| 9.2.3 Interim Data Analysis | 70 |
| CHAPTER 10: DATA COLLECTION AND MONITORING | 71 |
| 10.1 Case Report Forms and Other Data Collection | 71 |
| 10.1.1 Central Genetics Auditor (CGA) | 71 |
| 10.1.2 Genetics Committee (GC) | 71 |
| 10.1.3 Reading Center (RC) | 71 |
| 10.2 Study Records Retention | 71 |
| 10.3 Quality Assurance and Monitoring | 72 |
| 10.4 Protocol Deviations | 72 |
| CHAPTER 11: ETHICS/PROTECTION OF HUMAN PARTICIPANTS | 74 |
| 11.1 Ethical Standard | |
| 11.2 Institutional Review Boards | |
| 11.3 Informed Consent Process | 74 |
| 11.3.1 Consent Procedures and Documentation | 74 |
| 11.3.2 Participant and Data Confidentiality | 74 |
| 11.3.3 Future Use of Data and Ocular Images | 75 |
| CHAPTER 12: REFERENCES | 76 |

## **LIST OF ABBREVIATIONS**

| ABBREVIATION | DEFINITION |
|---|---|
| ADRP | Autosomal Dominant Retinitis Pigmentosa |
| AE | Adverse Event |
| BCVA | Best Corrected Visual Acuity |
| BRVT | Berkeley Rudimentary Vision Test |
| CC | Coordinating Center |
| CFR | Code of Federal Regulations |
| CGA | Central Genetics Auditor |
| CI | Confidence Interval |
| CME | Cystoid Macular Edema |
| CRF | Case Report Form |
| DHA | Docosahexaenoic Acid |
| EC | Ethics Committee |
| eCRF | Electronic Case Report Form |
| ERG | Electroretinogram |
| ETDRS | Early Treatment of Diabetic Retinopathy Study |
| EVA | Electronic Visual Acuity |
| EZ | Ellipsoid Zone |
| FAF | Fundus Autofluorescence |
| FDA | Food and Drug Administration |
| FFB | Foundation Fighting Blindness |
| ffERG | Full-field Electroretinogram |
| FST | Full-field Stimulus Threshold |
| GC | Genetics Committee |
| GCP | Good Clinical Practice |
| HOV | Hill of Vision |
| HRPP | Human Research Protection Program |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use |
| IOP | Intraocular Pressure |
| IRB | Institutional Review Board |
| IRD | Inherited Retinal Degeneration |
| KP | Kinetic Perimetry |
| LAR | Legally Authorized Representative |
| LLVA | Low Luminance Visual Acuity |
| LVP-FVQ II | L.V. Prasad-Functional Vision Questionnaire |

| ABBREVIATION | DEFINITION |
|---|---|
| MedDRA | Medical Dictionary for Regulatory Activities |
| MP | Microperimetry |
| MRDQ | Michigan Retinal Degeneration Questionnaire |
| N | Number or Sample Size |
| OCT | Optical Coherence Tomography |
| OD | Right Eye |
| OS | Left Eye |
| OU | Both Eyes |
| PHI | Protected Health Information |
| PI | Principal Investigator |
| PRO | Patient Reported Outcome |
| PROMIS®-29 | Patient-Reported Outcomes Measurement Information System |
| QA | Quality Assurance |
| QC | Quality Control |
| r | Pearson Correlation Coefficient |
| RC | Reading Center |
| RD | Retinal Dystrophy |
| RBM | Risk-Based Monitoring |
| RP | Retinitis Pigmentosa |
| RUSH2A | Rate of Progression in USH2A Related Retinal Degeneration Study |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SD-OCT | Spectral Domain Optical Coherence Tomography |
| SP | Static Perimetry |
| ULV-VFQ-50 | Ultra Low Vision-Visual Functioning Questionnaire |
| VA | Visual Acuity |
| VF | Visual Field |
| ViSIO-PRO | Visual Symptom and Impact Outcomes-Patient Reported Outcome |
| ViSIO-ObsRO | Visual Symptom and Impact Outcomes-Observer Reported Outcome |
| V <sub>tot</sub> | Total Volume |
| VUS | Variant(s) of Unknown Significance |
| YAC | Younger Age Cohort |
| α | Type I Error |

## PROTOCOL OUTLINE

| CATEGORY | DESCRIPTION |
|---|---|
| Title | Universal Rare Gene Study: A Registry and Natural History Study of Retinal Dystrophies Associated with Rare Disease-Causing Genetic Variants |
| Abbreviated<br>Name | Uni-Rare |
| Number of<br>Sites | Approximately 40 |
| Study Design | There are two components of this international, multicenter study: Registry A standardized genetic screening and a prospective, standardized, cross-sectional clinical data collection Enrollment is open to all genes on the RD Rare Gene List |
| | <ul> <li>Natural History Study</li> <li>A prospective, standardized, longitudinal Natural History Study</li> <li>Enrollment opens gene-by-gene, based on funding and within-gene Registry enrollment</li> </ul> |
| Objectives | The study objectives are as follows. See section 1.3 for details. Registry Objectives 1. Genotype Characterization 2. Cross-Sectional Phenotype Characterization (within gene) 3. Establish a Link to My Retina Tracker Registry (MRTR) 4. Ancillary Exploratory Studies – Pooling of Genes |
| | Natural History Study Objectives 1. Natural History (within gene) 2. Structure-Function Relationship (within gene) 3. Risk Factors for Progression (within gene) 4. Ancillary Exploratory Studies – Pooling of Genes |
| Précis | The <u>Registry</u> will establish genetically and clinically well-characterized cohorts of patients across hundreds of genetic variants associated with retinal dystrophy (RD). Characterization of these patients will accelerate eligibility screening for the Natural History Study, provide cross-sectional data on phenotype-genotype associations, and contribute to our knowledge of pathogenicity of these rare disease-causing variants. The <u>Natural History Study</u> will accelerate the identification and development of sensitive, reliable outcome measures for clinical trials, which will facilitate development of treatments for |
| | retinal dystrophies due to disease-causing genetic variants. The expected impact of the Natural History Study is as follows: 1. Describe the natural history of retinal degeneration in patients with rare disease-causing genetic variants 2. Identify sensitive structural and functional outcome measures to use for future multicenter clinical trials of rare inherited retinal degeneration |

| CATEGORY | DESCRIPTION | | |
|---|---|---|---|
| | 3. Identify well-defined subpopulations for future clinical trials of investigative treatments for rare inherited retinal degeneration | | |
| Participant<br>Duration | <ul> <li>Registry</li> <li>Registry/Screening Visit: Approximately 1-90 days</li> <li>Genetic screening: Approximately 30 days</li> <li>Annual phone calls: Up to approximately 48 months (or until gene is moved to the Natural History Study)</li> </ul> Natural History Study | | |
| Younger Age<br>Cohort | <ul> <li>Baseline Visit to 48-Month Follow-up Visit: Approximately 48 Months</li> <li>Participants ages ≥ 4 years and &lt; 8 years old will be designated as the Younger Age Cohort.</li> <li>Participants in this cohort will not be assigned a Vision Cohort.</li> <li>Registry/Screening Visit and Natural History Study Visits will have an abbreviated testing schedule, detailed in the Schedule of Study Visits and Procedures table.</li> </ul> | | |
| Without Colombia | | VF diameter ≥10° in VF diameter <10° in | |
| Vision Cohorts | 20/90 ou hotton | every meridian | any meridian |
| | 20/80 or better | Vision Cohort 1 | Vision Cohort 2 |
| | 20/100-20/400 | Vision Cohort 2 | Vision Cohort 2 |
| Protocol<br>Overview | The protocol overview is as follows. Also see flow charts in next section. 1. Screening Phase O Review patient's current genetic report* as having at least one gene on the RD Rare Gene List meeting one of the eligible Genetic Screening Criteria and review other eligibility criteria that can be evaluated based on medical history. O Complete Registry informed consent procedures according to overseeing Institutional Review Board (IRB)/Ethics Committee (EC) requirements. O Obtain ID on study website to be enrolled into initial screening. Complete the Registry/Screening Visit i. Confirm Registry eligibility criteria ii. Determine Vision Cohort** iii. Confirm Genetic Screening Criteria iv. Complete Registry data collection as part of the Registry/Screening Visit v. Participants meeting eligibility criteria to continue will be enrolled into the genetic screening phase *Genetic testing will not be performed in this study. A prior conclusive genetic test will be assessed for screening analysis. **Participants in the Younger Age Cohort will not be assigned a Vision Cohort. | | |

| CATEGORY | DESCRIPTION |
|---|---|
| CHILGORI | 2. Genetic Screening Phase |
| | o Genetic reports* for participants <i>enrolled into the genetic screening phase</i> will be uploaded to study website for review and confirmation by Central Genetics Auditor (CGA) as meeting <b>Genetic Screening Criteria</b> . |
| | <ul> <li>Participants confirmed as meeting those criteria will be considered <i>enrolled into</i><br/>the Registry.</li> </ul> |
| | *Genetic testing will not be performed in this study. A prior conclusive genetic test will be assessed for screening analysis. |
| | 3. Registry Phase |
| | <ul> <li>The flow of participants who are <i>enrolled into the Registry</i> depends on whether<br/>their causal gene is designated as a Natural History Study (NHS) Target Gene:</li> </ul> |
| | Not designated as NHS Target Gene: Annual phone calls up to 48 months from the Registry/Screening Visit or until gene is designated as NHS Target Gene. |
| | <ul> <li>Designated as NHS Target Gene: Participants will be considered<br/>pending enrollment into the NHS.</li> </ul> |
| | 4. Natural History Study (NHS) Phase |
| | o Participants <i>pending enrollment into the NHS</i> will do the following: |
| | i. Return to the clinic for the NHS Enrollment/Baseline Visit |
| | <ol> <li>Complete NHS informed consent procedures according to<br/>overseeing Institutional Review Board (IRB)/Ethics Committee<br/>(EC) requirements</li> </ol> |
| | 2. Confirm NHS eligibility criteria |
| | 3. Complete Baseline testing |
| | 4. Participants completing these steps will be considered <i>enrolled into the NHS</i> |
| | <ol> <li>Return to the clinic for follow-up visits according to Cohort<br/>specifications.</li> </ol> |
| | 1. Participants in the Younger Age Cohort and Vision Cohorts 1 and 2 will return to the clinic at 12, 24, 36 and 48 months from the Baseline Visit date for follow-up visits. |
| | 2. Participants in Vision Cohort 3 will have phone calls at 12, 24 and 36 months from the Baseline Visit date, and a study visit at 48 months. |
| | iii. After the 48-month follow-up visit, participation in the study will be completed for participants in all cohorts. |

| comes | <b>Functional Outcomes:</b> | | | | |
|---|---|---|---|---|---|
| | Key Assessments | Test | Equipment | Reading<br>Center | Registry (R)<br>or Natural<br>History Study<br>(NHS) |
| | Visual field sensitivity<br>measured with quantitative<br>topographic analysis (hill of<br>vision [HOV]) | Static Perimetry<br>(SP) | Octopus 900 Pro | Yes | R, NHS |
| | Early Treatment of Diabetic<br>Retinopathy Study<br>(ETDRS) / HOTV Best<br>Corrected Visual Acuity<br>(BCVA) letter score | Visual Acuity (VA) | Electronic Visual Acuity (EVA) system or ETDRS/HOTV charts | N/A | R, NHS |
| | Low visual acuity test – for participants unable to see ETDRS letters | Low Visual Acuity | Berkeley<br>Rudimentary<br>Vision Test<br>(BRVT) | N/A | R, NHS |
| | ETDRS/HOTV best corrected low luminance visual acuity letter score | Low Luminance<br>Visual Acuity<br>(LLVA) | Electronic Visual<br>Acuity (EVA)<br>system or<br>ETDRS/HOTV<br>charts | N/A | R, NHS |
| | Mean retinal sensitivity | Fundus guided<br>Microperimetry<br>(MP) | MAIA | Yes | NHS |
| | Contrast sensitivity function | Contrast sensitivity | CSV-1000E chart | N/A | NHS |
| | Retinal function using amplitudes and timing in response to rod- and conespecific stimuli | Full-field<br>Electroretinogram<br>(ffERG) | Diagnosys Espion | No | NHS |
| | Full-field retinal sensitivity | Full-field stimulus<br>threshold (FST)<br>testing to blue,<br>white, and red<br>stimuli | Diagnosys Espion | No | NHS |
| | Color vision function | Color vision | Lanthony D15 | N/A | NHS |
| | Structural Outcomes: | | | | |
| | Key Assessments | Test | Equipment | Reading<br>Center | Registry (R)<br>or Natural<br>History Study<br>(NHS) |
| | Ellipsoid zone (EZ) area;<br>outer nuclear layer and<br>ganglion cell layer<br>thicknesses | Spectral Domain<br>Optical Coherence<br>Tomography (SD-<br>OCT) | Heidelberg<br>Spectralis | Yes | R, NHS |

| | Qualitative and quantitative assessments of autofluorescence pattern | Fundus<br>Autofluorescence<br>(FAF) | Optos | Yes | NHS |
|---|---|---|---|---|---|
| | Patient Reported Outcomes (PROs) (NHS only): | | | | |
| | Adults 18 years or older | at Baseline: | | | |
| | o Michigan Retinal De | egeneration Questions | naire (MRDQ) | | |
| | <ul> <li>Patient-Reported Outcomes Measurement Information System (PROMIS®-29)</li> <li>Visual Symptom and Impact Outcomes-Patient Reported Outcome (ViSIO-PRO)</li> <li>Ultra Low Vision-Visual Functioning Questionnaire (ULV-VFQ-50) – Vision Cohort 3 only</li> </ul> | | | | |
| | Adolescents 12-17 years | at Baseline: | | | |
| | <ul> <li>Visual Symptom and Impact Outcomes-Patient Reported Outcome (ViSIO-PRO)</li> <li>L. V. Prasad-Functional Vision Questionnaire (LVP-FVQ II)</li> </ul> | | | | |
| | • Children 8-11 years at Baseline: | | | | |
| | <ul> <li>Visual Symptom and Impact Outcomes-Observer Reported Outcome (ViSIO-ObsRO)</li> <li>L. V. Prasad-Functional Vision Questionnaire (LVP-FVQ II)</li> </ul> | | | | |
| | Children 4-7 years at Ba Visual Symptom and | <u>seline</u> :<br>d Impact Outcomes-C | bserver Reported | Outcome (V | /iSIO-ObsRO) |
| RD Rare Gene<br>List | The RD Rare Gene List for the Uni-Rare study (see Uni-Rare Clinical Site Manual of Procedures) represents all known genes for which variants may be associated with retinal dystrophy (RD) and have not already been studied in a trial at the time this protocol was finalized. | | | | |
| Population | Key Eligibility Criteria – Determined at the Registry/Screening Visit | | | | |
| • | The entire list of eligibility criteria in protocol section 2.4.1 must be reviewed at the Registry/Screening Visit. Participants meeting eligibility criteria will continue to <i>enroll into the genetic screening phase</i> . | | | | |
| | A key subset of the eligibilit | y criteria includes the | following: | | |
| | • Age ≥ 4 years of age | 2 | | | |
| | Clinical diagnosis of retinal dystrophy (RD) | | | | |
| | <ul> <li>Must have a gene on the RD Rare Gene List which meets one of the following Genetic<br/>Screening Criteria*</li> </ul> | | | | |
| | <ul> <li>Inheritance Pattern is Recessive <u>and</u> has at least 2 disease-causing variants which<br/>are homozygous or heterozygous <i>in trans</i></li> </ul> | | | | |
| | <u>OR</u> | | | | |
| | phase <u>and</u> n | Pattern is Recessive <u>a</u> neets all the following segregation in trans: | | - | |
| | 1. Inve | estigator confirms gen<br>osomal recessive inher | | pe are cons | istent with |
| | | 2 disease-causing values | riants have <u>not</u> bee | en reported | in cis in variant |

- 3. <u>No</u> additional potentially pathogenic variants were found on the gene (and the sequencing data for the gene were sufficiently robust to detect any additional potentially pathogenic variants)
- 4. <u>No</u> potentially pathogenic variants were found in other common, likely candidate genes for the proposed condition

#### <u>OR</u>

o Inheritance Pattern is Dominant, X-linked, or Mitochondrial <u>and</u> has at least 1 disease-causing variant

\*Based on prior conclusive genetic report from a clinically certified lab (or from a research lab that has been approved by the study Genetics Committee).

#### **Genetic Screening Phase**

The Genetic Screening Phase will confirm genetic cause of disease via final Central Genetics Auditor (CGA) review for all participants.

#### **Registry Cohort Criteria**

At the end of the Genetic Screening Phase the following must be documented to be eligible to *enroll into the Registry*:

Participant's genetic cause of disease has been confirmed by Central Genetics Auditor (CGA) as meeting one of the **Genetic Screening Criteria** for a gene on the **RD Rare Gene List**.

#### **Natural History Study Cohort Criteria**

Participants who meet the final *Registry Cohort Criteria* will be eligible to enroll into the NHS <u>if</u> and when their causal gene is designated as an NHS Target Gene. This gene-by-gene designation will be made by the Executive Committee on an ongoing basis and may depend on funding resources as well as Registry enrollment numbers within gene. NHS consent will be required, and additional NHS eligibility criteria will be confirmed prior to enrollment into the NHS.

#### Sample Size

#### Registry

- Recruitment will continue until 1,500 participants meet the final *Registry Cohort Criteria*, unless the Executive Committee terminates recruitment due to feasibility.
- A maximum of 150 participants in Vision Cohort 3.
- A maximum of 100 participants where Inheritance Pattern is Recessive and phase is unknown.
- A maximum of 100 participants within gene.

The Executive Committee will monitor enrollment distributions across genes, inheritance patterns, vision cohorts, and age cohorts with the planned caps as noted. Enrollment in some genes, inheritance patterns, vision cohorts, or age cohorts may be encouraged to ensure appropriate representation, and some caps may be adjusted if needed.

#### **Natural History Study**

• The Natural History Study sample size for each gene will depend on the Registry enrollment; a maximum of 100 participants within gene.

#### FLOW CHART – SCREENING PHASE

## Screening Phase

#### **Initial Enrollment**

- Investigator reviews patient's genetic report as having at least one gene on the RD Rare Gene List meeting Genetic Screening Criteria and reviews other eligibility criteria that can be evaluated based on medical history
- Consent participant according to overseeing IRB/Ethics Committee requirements
- Obtain ID on study website

Participant is "Enrolled into the initial screening"

### Registry/Screening Visit

See Schedule of Study Visits and Procedures

- Eligibility Criteria Assessment
- Demographics
- Medical History
- Ocular Exam
- Visual Acuity (incl. refraction and LLVA/BRVT as needed)\*
- Intraocular Pressure
- SD-OCT\*
- Static Perimetry\*
- Kinetic visual field III4e\* (performed within last 18 months)
- Determination of Vision Cohort\*
- Genetic Screening Criteria assessment

If determined not eligible at any step:

Discontinue Screening Visit; Participant is "Initial screen failure"



If eligible:

Participant is "Enrolled into genetic screening phase"

\* Testing not performed

in Younger Age Cohort

**Begin Genetic Screening Phase** 

#### Genetic Screening Criteria

To enter the Genetic Screening Phase, participants must have a gene on the **RD Rare Gene List** meeting one of the following:

| the following. | |
|---|---|
| Inheritance Pattern <sup>1</sup> | Variant Documentation <sup>2</sup> |
| Recessive | At least 2 disease-causing variants which are homozygous or heterozygous in trans |
| | <u>OR</u> |
| | 2 disease-causing variants with unknown phase <u>and</u> meets all the following additional informatic criteria |
| | that is consistent with likely segregation in trans |
| | Investigator confirms genotype and phenotype are consistent with autosomal recessive |
| | inheritance |
| | The 2 disease-causing variants have <u>not</u> been reported in cis in variant databases |
| | <ul> <li>No additional potentially pathogenic variants were found on the gene (and the sequencing data</li> </ul> |
| | for the gene were sufficiently robust to detect any additional potentially pathogenic variants) |
| | <ul> <li>No potentially pathogenic variants were found in other common, likely candidate genes for the</li> </ul> |
| | proposed condition |
| Dominant, X-linked, | At least 1 disease-causing variant |
| or Mitochondrial | |

- 1- Based on protocol-defined RD Rare Gene List mapping.
- 2- Based on prior conclusive genetic report from a clinically certified lab (or from a research lab that has been approved by the study Genetics Committee).

## FLOW CHART – GENETIC SCREENING PHASE



#### Final Registry Cohort Criteria

Participant's genetic cause of disease has been <u>confirmed by CGA</u>\* as meeting one of the following, for a gene on the RD Rare Gene List:

 Inheritance Pattern is Recessive <u>and</u> has at least 2 disease-causing variants which are homozygous or heterozygous in trans

#### OR

- Inheritance Pattern is Recessive <u>and</u> has 2 disease-causing variants with unknown phase <u>and</u> meets all the following additional informatic criteria that is consistent with likely segregation *in trans* 
  - > Investigator confirms genotype and phenotype are consistent with autosomal recessive inheritance
  - ➤ The 2 disease-causing variants have <u>not</u> been reported *in cis* in variant databases
  - No additional potentially pathogenic variants were found on the gene (and the sequencing data for the gene were sufficiently robust to detect any additional potentially pathogenic variants)
  - No potentially pathogenic variants were found in other common, likely candidate genes for the proposed condition

#### <u>OR</u>

• Inheritance Pattern is Dominant, X-linked, or Mitochondrial and has at least 1 disease-causing variant

\*Based on prior conclusive genetic report from a clinically certified lab (or from a research lab that has been approved by the study Genetics Committee).

Periodically, all genetic reports of participants enrolled into the final registry cohort will be evaluated by the Genetics Committee for the following. This analysis will not change eligibility to be enrolled into the final registry cohort.

- Interpretation of pathogenicity
- · Genetic classifications for analyses

## FLOW CHART - REGISTRY PHASE



## FLOW CHART - NATURAL HISTORY STUDY



## SUMMARY OF PROCEDURES FOR THE REGISTRY/SCREENING VISIT, GENETIC SCREENING PHASE, AND REGISTRY PHASE

| Visit/Phase | Registry/<br>Screening | Genetic<br>Screening | 12M | 24M | 36M | 48M |
|---|---|---|---|---|---|---|
| VISITI HASC | Visit | Phase | 12111 | 27111 | 30111 | 401VI |
| Phone Call Target Windows <sup>a</sup> | | | Wk<br>52 ± 8 | Wk<br>104 ± 8 | Wk<br>156 ± 8 | $Wk \\ 208 \pm 8$ |
| Participant-Level Procedures | | | | | | |
| Registry Informed Consent | X | | | | | |
| Collect MyRetinaTrackerID (if participating and consented to provide) | X | | | | | |
| Eligibility Criteria Assessment | X | | | | | |
| Demographics | X | | | | | |
| Medical History (incl. pre-existing conditions, symptomology history, medications) | X | | | | | |
| Genetic Report Assessment (incl. Genetic Screening Criteria) | X | | | | | |
| Determination of Vision Cohort ° | X | | | | | |
| CGA Confirmation of Genetic Cause of Disease and Final Genetic Eligibility | | X | | | | |
| Phone Call (patient contact only; no data collection) | | | X | X | X | X |
| Ocular Procedures b – all testing performed in each eye | | | | | | |
| Complete Ophthalmic Exam <sup>d</sup> | X | | | | | |
| Visual Acuity (EVA preferred or ETDRS charts); with refraction and LLVA/BRVT ° | X | | | | | |
| Intraocular Pressure <sup>e</sup> | X | | | | | |
| SD-OCT Volume Scans <sup>c</sup> (Heidelberg Spectralis) | X | | | | | |
| SD-OCT Vertical and Horizontal Scans <sup>c</sup> (Heidelberg Spectralis) | X | | | | | |
| Static Perimetry <sup>c</sup> (Octopus 900 Pro) | X | | | | | |
| Kinetic VF III4e c, f (Kinetic Perimetry) | X | | | | | |

- a. Timed from Registry/Screening Visit; annually up to four (4) years <u>or</u> until participant's gene is designated as an NHS Target Gene.
- b. The Registry/Screening Visit date is defined as the start date of all Registry/Screening testing. All Registry/Screening testing must be completed within ninety (90) days of the Registry/Screening Visit date (except for ophthalmic exam and kinetic VF, as noted in <u>d</u> and <u>f</u> below). *All procedures are considered standard care.*
- c. Testing not performed in Younger Age Cohort.
- d. Ophthalmic exam can be performed at Registry/Screening Visit, or a historical measurement performed within the last six (6) months prior to the Registry/Screening Visit. The ophthalmic exam includes slit-lamp biomicroscopy and indirect ophthalmoscopy.
- e. Intraocular pressure (IOP) measurements are to be taken prior to pupil dilation.
- f. Vision Cohort 1 and 2: Historical measurement performed within the last eighteen (18) months prior to the Registry/Screening Visit. If a historical measurement is not available, then perform the Kinetic VF III4e at the Registry/Screening Visit. Vision Cohort 3: Collect the most recent historical measurement prior to the Registry/Screening Visit, if available. Kinetic VF III4e does not need to be performed at screening if a historical measurement is not available.

## SCHEDULE OF STUDY VISITS AND PROCEDURES FOR THE NATURAL HISTORY STUDY: <u>Younger Age Cohort</u>

| Visit | Baseline a | 12M <sup>b</sup> | 24M <sup>b</sup> | 36M <sup>b</sup> | <b>48M</b> <sup>b</sup> |
|---|---|---|---|---|---|
| Target Windows | (Day 0) | Wk<br>52 ± 4 | $\begin{array}{c} Wk \\ 104 \pm 4 \end{array}$ | Wk<br>156 ± 4 | Wk<br>208 ± 4 |
| Participant-Level Procedures | | | | | |
| NHS Informed Consent | X | | | | |
| Eligibility Criteria Assessment | X | | | | |
| Concomitant Medications / Adverse Events / Medical History Update | X | X | X | X | X |
| Patient Reported Outcomes (PROs) | X | | X | | X |
| Ocular Procedures – all testing performed in each eye | | | | | |
| Complete Ophthalmic Exam <sup>c</sup> | X | X | X | X | X |
| Visual Acuity (HOTV); with refraction and LLVA/BRVT | X | X | X | X | X |
| Intraocular Pressure d | X | X | X | X | X |
| Color Vision (Lanthony D15) | X | X | X | X | X |
| SD-OCT Volume Scans (Heidelberg Spectralis e) | X | X | X | X | X |
| SD-OCT Vertical and Horizontal Scans (Heidelberg Spectralis <sup>e</sup> ) | X | X | X | X | X |
| Axial Length and Corneal Curvature Measurements | X | X | X | X | X |
| Optos Color Photos h | X | | | | |
| Optos Fundus Autofluorescence h | X | X | X | X | X |
| Full-field ERG (Diagnosys Espion) f, h | X | | | | X |
| Full-field Stimulus Threshold (Diagnosys Espion) h | X | X | X | X | X |
| Age-Up Procedures <sup>g</sup> – for participants who turn 8 y/o during study period | | | | | |
| Static Perimetry (Octopus 900 Pro) | | X | X | X | X |
| Fundus Guided Microperimetry (MAIA) h | | X | X | X | X |
| Contrast Sensitivity (CSV-1000E) | | X | X | X | X |

- a. Baseline testing must be started within seven (7) days of NHS eligibility confirmation. The Baseline Visit date is defined as the start date of all Baseline testing. All Baseline testing must be completed within thirty (30) days of the Baseline Visit date, with the following exceptions:
  - If the Baseline Visit date is within 3 months of the Registry/Screening Visit testing date for the ophthalmic exam or IOP exam, the testing performed as part of the Registry/Screening Visit for these modalities may be used for the Baseline Visit.
  - PROs may be completed in person or remotely any time within 6 months after Baseline Visit date.
- b. All NHS Follow-up Visit testing must be completed on the same day, with the following exception:
  - PROs may be completed in person or remotely any time within the Allowable Window of the associated visit.
- c. Ophthalmic exam includes slit-lamp biomicroscopy and indirect ophthalmoscopy. It is recommended that the ocular exam is completed at approximately the same time of day at each visit using the same equipment.
- d. Intraocular pressure (IOP) measurements are to be taken prior to pupil dilation.
- e. If a Younger Age Cohort participant is unable to perform OCT testing on the Heidelberg Spectralis, the handheld Bioptogen/Envisu may be used to perform OCT testing for qualitative purposes with approval from the Coordinating Center.
- f. If ERG has been undetectable in the past, there is no need to perform at Baseline Visit; if ERG is undetectable at Baseline Visit, there is no need to perform at 48M at the investigator's discretion.
- g. Participants in the Younger Age Cohort who turn 8 years old (age-up) during the NHS study period should attempt to have static perimetry, microperimetry, and contrast sensitivity testing performed at the next study visit after they turn 8 years old and at every subsequent visit, until the end of the study period.
- h. If a site does not have the required equipment, participation in this test may be waived with approval from the Coordinating Center.

## SCHEDULE OF STUDY VISITS AND PROCEDURES FOR THE NATURAL HISTORY STUDY: <u>VISION COHORTS 1 AND 2</u>

| Visit | Baseline a | 12M <sup>b</sup> | <b>24M</b> <sup>b</sup> | <b>36M</b> <sup>b</sup> | <b>48M</b> <sup>b</sup> |
|---|---|---|---|---|---|
| Visit Target Windows | (Day 0) | Wk<br>52 ± 4 | Wk<br>104± 4 | Wk<br>156± 4 | Wk<br>208± 4 |
| Participant-Level Procedures | | | | | |
| NHS Informed Consent | X | | | | |
| Eligibility Criteria Assessment | X | | | | |
| Concomitant Medications / Adverse Events / Medical History Update | X | X | X | X | X |
| Patient Reported Outcomes (PROs) | X | | X | | X |
| Ocular Procedures – all testing performed in each eye | • | | | | |
| Complete Ophthalmic Exam <sup>c</sup> | X | X | X | X | X |
| Visual Acuity (EVA preferred or ETDRS charts); with refraction and LLVA/BRVT | X | X | X | X | X |
| Intraocular Pressure d | X | X | X | X | X |
| Color Vision (Lanthony D15) | X | X | X | X | X |
| Contrast Sensitivity (CSV-1000E) | X | X | X | X | X |
| SD-OCT Volume Scans (Heidelberg Spectralis) | X | X | X | X | X |
| SD-OCT Vertical and Horizontal Scans (Heidelberg Spectralis) | X | X | X | X | X |
| Axial Length and Corneal Curvature Measurements <sup>e</sup> | X | X | X | X | X |
| Optos Color Photo <sup>h</sup> | X | | | | |
| Optos Fundus Autofluorescence h | X | X | X | X | X |
| Full-field ERG (Diagnosys Espion) f, h | X | | | | X |
| Full-field Stimulus Threshold (Diagnosys Espion) h | X | X | X | X | X |
| Static Perimetry (Octopus 900 Pro) <sup>g</sup> | X | X | X | X | X |
| Fundus Guided Microperimetry (MAIA) <sup>g, h</sup> | X | X | X | X | X |

- a. Baseline testing must be started within seven (7) days of eligibility confirmation. Baseline Visit date is defined as the start date of all Baseline testing. All Baseline testing must be completed within thirty (30) days of the Baseline Visit date, with the following exceptions:
  - If the Baseline Visit date is within 3 months of the Registry/Screening Visit testing date for the visual acuity (VA), static perimetry, SD-OCT (volume and V/H), ophthalmic exam or IOP exams, the testing performed as part of the Registry/Screening Visit may be used for the Baseline Visit. A second static perimetry test would still need to be performed at the Baseline Visit, as noted in helow.
  - PROs may be completed in person or remotely any time within 6 months after Baseline Visit date.
- b. All NHS Follow-up Visit testing must be completed on the same day, with the following exception:
  - PROs may be completed in person or remotely any time within the Allowable Window of the associated visit.
- c. Ophthalmic exam includes slit-lamp biomicroscopy and indirect ophthalmoscopy. It is recommended that the ocular exam be completed at approximately the same time of day at each visit using the same equipment.
- d. Intraocular pressure (IOP) measurements are to be taken prior to pupil dilation.
- e. Axial length and corneal curvature measurements will be completed at the Baseline Visit for all participants. Only individuals who are under 18 years old at the Baseline Visit will continue to have measurements taken at every annual visit until study completion.
- f. If ERG has been undetectable in the past, there is no need to perform at Baseline Visit; if ERG is undetectable at Baseline Visit, there is no need to perform at 48M at the investigator's discretion.

| g. | For static perimetry and microperimetry, all participants will complete two tests for the Baseline Visit. The |
|---|---|
| | results will be compared according to the visual field criteria in section 4.3.2 to determine if a third test is |
| | needed |

h. If a site does not have the required equipment, participation in this test may be waived with approval from the Coordinating Center.

## SCHEDULE OF STUDY VISITS AND PROCEDURES FOR THE NATURAL HISTORY STUDY: <u>VISION COHORT 3</u>

| Visit | Baseline a | 12M | 24M | 36M | <b>48M</b> <sup>b</sup> |
|---|---|---|---|---|---|
| Target Windows | (Day 0) | $Wk$ $52 \pm 4$ (Phone call only) | Wk<br>104±4<br>(Phone call<br>only) | Wk<br>156± 4<br>(Phone call<br>only) | Wk<br>208± 4 |
| Participant-Level Procedures | | | | | |
| NHS Informed Consent | X | | | | |
| Eligibility Criteria Assessment | X | | | | |
| Concomitant Medications / Adverse Events / Medical History Update | X | X | X | X | X |
| Patient Reported Outcomes (PROs) | X | | | | X |
| Ocular Procedures – all testing performed in each eye | | | | | |
| Complete Ophthalmic Exam <sup>c</sup> | X | | | | X |
| Visual Acuity (EVA preferred or ETDRS charts); with refraction and LLVA/BRVT | X | | | | X |
| Intraocular Pressure d | X | | | | X |
| SD-OCT Volume Scans (Heidelberg Spectralis) | X | | | | X |
| SD-OCT Vertical and Horizontal Scans (Heidelberg Spectralis) | X | | | | X |
| Axial Length and Corneal Curvature Measurements e | X | | | | X |
| Optos Color Photos <sup>f</sup> | X | | | | |
| Optos Fundus Autofluorescence <sup>f</sup> | X | | | | X |
| Full-field Stimulus Threshold (Diagnosys Espion) f | X | | | | X |

- a. Baseline testing must be started within seven (7) days of eligibility confirmation. Baseline Visit date is defined as the start date of all Baseline testing. All Baseline testing must be completed within thirty (30) days of the Baseline Visit date, with the following exceptions:
  - If the Baseline Visit date is within 3 months of the Registry/Screening Visit testing date for the visual acuity (VA), SD-OCT (volume and V/H), ophthalmic exam or IOP exams, the testing performed as part of the Registry/Screening Visit may be used for the Baseline Visit.
  - PROs may be completed in person or remotely any time within 6 months after Baseline Visit date.
- b. All NHS Follow-up Visit testing must be completed on the same day, with the following exception:
  - PROs may be completed in person or remotely any time within the Allowable Window of the associated visit.
- c. Ophthalmic exam includes slit-lamp biomicroscopy and indirect ophthalmoscopy. It is recommended that the ocular exam is completed at approximately the same time of day at each visit using the same equipment.
- d. Intraocular pressure (IOP) measurements are to be taken prior to pupil dilation.
- e. Axial length and corneal curvature measurements will be completed at the Baseline Visit for all participants. Only individuals who were under 18 years old at the Baseline Visit will also have measurements taken at the 48M visit.
- f. If a site does not have the required equipment, participation in this test may be waived with approval from the Coordinating Center

## **Chapter 1: Background Information**

#### 1.1 Introduction

1

2

- 3 Inherited retinal degenerations (IRDs) affect approximately 2 to 3 million people worldwide.<sup>1</sup>
- 4 The rise of promising treatment approaches has increased rapidly in recent years, include gene
- 5 editing and augmentation (early-stage disease), neuroprotection (mid-stage disease), prosthetics,
- optogenetics, and cell therapy to restore some light sensation (late-stage disease). 1,2 Despite
- advancements in therapy development, and a growing number of interventional trials
- 8 (https://www.clinicaltrials.gov/) for IRDs, there remain significant hurdles to designing trials and
- 9 moving therapy through the development process. Several papers have reviewed unmet needs
- and identified top priorities to move the promise of treatment forward amongst a complex
- landscape of IRD research.<sup>3-7</sup> The common theme among the recommendations is the vital need
- for natural history studies, the foundational basis for trial design and drug development. The
- following sections summarize the key gaps in IRD research that natural history studies can
- 14 address.

15

#### 1.1.1 Identifying Optimal IRD Patient Populations for Target Therapies

- 16 IRDs are genetically diverse (280 causative genes have been identified to date)
- 17 (<a href="https://sph.uth.edu/retnet/">https://sph.uth.edu/retnet/</a>) and have vastly different clinical manifestations, including age of
- onset, severity of disease, rate of progression, and structural and functional abnormalities.
- 19 Understanding this phenotypic heterogeneity is a major challenge for potential therapy
- developers. It is critical to identify genetic factors impacting disease severity and progression,
- 21 including the impact of mutation-specific variations within genes. Natural history data, both
- longitudinal and cross-sectional, within each gene population is needed to understand these
- 23 differences, and ideally these studies would include enough cases to evaluate a variety of
- subgroups across genetic, phenotypic, and environmental factors.<sup>3-7</sup>

### 1.1.2 Develop and Validate Outcome Measures for Progression of IRDs

- The cornerstone of good trial design is a good endpoint. Identifying the best candidate endpoint
- 27 for evaluating progression of disease, and ultimately treatment effects in a trial, requires
- 28 consideration of many properties. These include sensitivity, reproducibility, correlation with
- other measures of disease progression, how much within-person change is beyond measurement
- variability, and whether within-person change is clinically meaningful. For a given treatment, the
- best measure also depends on the expected benefit; restoration of vision versus slowing of
- progression. Since IRDs are genetically diverse, understanding these properties within each gene
- 33 is important.<sup>3-7</sup>
- 34

25

- The list of candidate endpoints to measure and understand IRD progression is vast. <u>Visual</u>
- 36 **function outcomes,** such as visual acuity (VA), contrast sensitivity, color vision, microperimetry
- 37 (MP), full-field stimulus threshold (FST) and full-field electroretinogram (ffERG), measure
- 38 performance of the components of the visual system in the clinical environment and represent the
- measures of what is clinically meaningful. **Structural or anatomical measures**, such as fundus
- autofluorescence (FAF) and optical coherence tomography (OCT), represent candidate
- biomarkers or surrogate endpoints that hold the potential to predict clinical benefit. Structural
- measures are an expanding area of IRD research due to new technologies and better imaging

- acquisition and interpretation techniques and is an area of priority identified by gap analyses.
- 44 Functional vision measures, which are designed to reflect real-life challenges in daily activities,
- include patient-reported outcomes. Although a variety of tools exist, little is known about their
- applicability within each genotype.<sup>3-7</sup>

47

54

62

63

72

- 48 A relatively small number of endpoints defined by these measures have been accepted by the
- 49 Food and Drug Administration (FDA) and other regulatory bodies to study therapeutic efficacy
- in IRD trials. The extreme genetic heterogeneity of IRDs and diversity of resulting disease
- 51 progression further complicates the decision of which endpoint to use for a given gene therapy
- 52 trial. Gene-specific natural history studies can provide longitudinal data to understand the
- 53 properties of these measures and facilitate development of appropriate endpoints for trial design.

#### 1.1.3 Other Gaps Addressed by Natural History Studies

- Natural history studies address numerous other challenges faced in clinical trial design and
- 56 implementation, including understanding the time course of disease progression (which informs
- 57 trial duration and testing schedule), evaluating demographic and epidemiological estimates of
- 58 prevalence and disease characteristics (which may be addressed by cross-sectional studies), and
- 59 identifying expert clinical centers with staff trained to follow standardized protocols. They also
- shed light on intangibles and unknowns, which ultimately saves resources, increases efficiencies,
- and improves quality of future interventional trials built upon these lessons learned.

#### 1.1.4 Unique Challenges in Ultra-Rare Genes

- Ultra-rare genes present a special challenge in addressing these knowledge gaps and represent a
- significant portion of IRD genes. Two hundred and forty-eight (248) genes out of three hundred
- and seventy-four (374) potential IRD genes listed in the FFB Consortium 2021 Gene Poll had
- less than twenty (20) patients counted as having retinal dystrophy (RD) linked to that causal
- 67 gene, across all thirty-two (32) sites reporting in the Poll (data not published). Small sample sizes
- create less precision around estimates and difficulty or inability to evaluate factors related to
- disease severity and progression or correlation among outcomes. Further study is needed to
- 70 identify similar disease mechanisms and whether there are methods by which researchers could
- 71 pool data across genes for these objectives.

#### 1.2 Rationale for a Universal Rare Gene Study

- Individual natural history studies for each rare RD gene are not feasible. Many centers have as
- few as one (1) two (2) patients for a particular RD gene and may not be able to devote
- 75 resources needed to implement each study. Individual studies also require considerable startup
- time (e.g., contracts, IRB/Ethics Committee approvals) and study management expenses
- regardless of the number of patients. A single, universal protocol under which all rare RD genes
- may be enrolled would address these inefficiencies.
- Because of the vast phenotypic diversity, simultaneous open enrollment of all rare RD genes
- directly into a longitudinal natural history study is problematic. Unfocused enrollment efforts
- spread across hundreds of genes will dilute timelines for data collection and analysis objectives
- within targeted genes. A solution is to create a universal registry open to all rare RD genes, to
- cross-sectionally characterize patients within all rare RD genes (mild, moderate, and severe
- vision loss) so they are ready to be enrolled into a subsequent universal longitudinal natural

| 85 | history | y study | as their gene is selected. This two-phase platform will (1) eliminate repetitive |
|---|---|---|---|
| 86 | proces | ses like | certification, training, regulatory approval, contract agreements, (2) reduce costs |
| 87 | and ac | celerate | e timelines for longitudinal studies and (3) leverage a large sample size and |
| 88 | | | data collection in the cross-sectional study to explore the extent to which genes with |
| 89 | | | hanisms of disease have similar clinical manifestations (e.g., determine if and how |
| 90 | | | nay be pooled in some analyses). |
| 91 | 1.3 St | udy Ob | jectives |
| 92 | Regist | try Obj | <u>ectives</u> |
| 93 | 1. | Genot | ype Characterization |
| 94 | | a. | Establish a database of patients completing a standardized genetic screening |
| 95 | | | process confirming retinal dystrophy is associated with disease-causing genetic |
| 96 | | | variants (and thereby confirmed genetically eligible for a potential <b>natural</b> |
| 97 | | | history study) |
| 98 | | b. | Evaluate characteristics of genetic variants |
| 99 | 2. | Cross | -Sectional Phenotype Characterization* |
| 100 | | a. | Characterize cross-sectional retinal dystrophy associated with disease-causing |
| 101 | | | genetic variants using functional and structural measures, within gene |
| 102 | | | i. Ideally where within-gene sample size is 20 or more |
| 103 | | b. | Structure-function relationships will also be explored within-gene |
| 104 | | | i. Ideally where within-gene sample size is 20 or more |
| 105 | | c. | Risk factors for disease severity will also be explored within-gene |
| 106 | | | i. Ideally where within-gene sample size is 40 or more |
| 107 | 3. | Estab | lish a Link to My Retina Tracker Registry (MRTR) |
| 108 | | a. | Register MRTR participants for exploratory analysis of data between registry |
| 109 | | | databases, as permissible within the scope of signed informed consent(s) |
| 110 | 4. | Ancill | ary Exploratory Studies - Pooling of Genes |
| 111 | | a. | Explore whether phenotype-genotype associations within biological mechanisms |
| 112 | | | or other factors (such as age or disease duration) will allow pooling of genes for |
| 113 | | | cross-sectional analysis objectives |
| 114 | | b. | If pooling is determined appropriate, evaluate objective 2 above within |
| 115 | | | appropriate pooling groups |
| 116 | | | |
| 117 | Natur | al Histo | ory Study Objectives |
| 118 | Within | n-Gene | Objectives* |
| 119 | The fo | llowing | g objectives will be evaluated within gene. |
| 120 | 1. | Natur | al History |
| 121 | | a. | Characterize the natural history of retinal degeneration associated with disease- |
| 122 | | | causing genetic variants over 4 years, using functional, structural, and patient- |
| 123 | | | reported outcome measures |
| 124 | | b. | Ideally where within-gene sample size is 20 or more |
| 125 | 2. | | ture-Function Relationship |
| 126 | | a. | Explore whether structural outcome measures can be validated as surrogates for |
| 127 | | | functional outcomes in individuals with disease-causing genetic variants |
| 128 | | b. | Ideally where within-gene sample size is 20 or more |

129

#### 3. Risk Factors for Progression 130

- Explore possible risk factors (genotype, phenotype, environmental, and comorbidities) for progression of the outcome measures at 4 years in individuals with disease-causing genetic variants
- b. Ideally where within-gene sample size is 40 or more

134 135 136

137

131

132

133

\*Applicability of within-gene objectives will depend on within-gene sample size as noted above. If less than 20, the primary objective will be limited to describing the cohort in the form of case histories. Objectives may still be explored depending on the needs of a specific gene.

138 139 140

141

142

143

144

145

146

147

156

157

158

159

160

161

162

163

164

165

166

167

168

### Across-Genes Objective

The following objective will be evaluated across genes.

## 4. Ancillary Exploratory Studies - Pooling of Genes

a. Explore whether phenotype-genotype associations within biological mechanisms or other factors (such as age or disease duration) will allow pooling of genes for longitudinal analysis objectives

#### 1.4 Potential Risks and Benefits

#### 1.4.1 Known Potential Risks

- Most examination procedures are considered part of standard care for retinal degenerations. This 148
- study will be capturing some information about participants that include identifiable, personal 149
- information, like date of birth (will be collected if permitted by site's regulatory bodies). The 150
- study has procedures in place to protect that information. However, there is a chance that a loss 151
- of that protection could occur. This would be a loss of confidentiality. There are special efforts 152
- being made to ensure that this does not happen. 153
- The sections below summarize the risks and discomforts that may be occur during the period of 154
- prospective data collection. 155
  - Risks associated with testing VA, KP, SP, MP, FST, ERG, OCT, and PROs may include boredom and frustration, but no lasting adverse effects are associated with these noninvasive tests
  - Dilating eye drops will be used as part of the ophthalmic examination and before some tests. Dilating eye drops may sting, cause light-sensitivity, or an allergic reaction. There is a small risk of inducing a narrow-angle glaucoma attack from the pupil dilation. However, all participants will have had prior pupil dilation usually on multiple occasions and therefore the risk is extremely small. If glaucoma occurs, treatment is available.
  - In rare instances, the cornea may be scratched during measurement of IOP or use of a contact lens electrode. An abrasion like this may be painful, but it heals quickly with no lasting effects. If a participant experiences a corneal abrasion, a tear ointment may be administered, and an eye patch or gauze may be placed over the eye.

#### 1.4.2 Known Potential Benefits

Study participants are not expected to benefit directly from participation in this study. Study 169 participants participating in this study may benefit from close attention from the study personnel 170

- and Investigator(s). The risks of participating in the study are outweighed by the benefits.
- Benefits include increased attention from the study personnel and the ability to contribute to
- increased understanding of the cross-sectional description and natural history of retinal
- degenerations due variants in rare genes, which may contribute to future development of
- treatments.

176

180

#### 1.4.3 Risk Assessment

- 177 The risk level for this protocol is considered no greater than minimal risk. A risk-based
- monitoring approach will be followed, consistent with the FDA "Guidance for Industry
- Oversight of Clinical Investigations A Risk-Based Approach to Monitoring" (August 2013).

#### 1.5 General Considerations

- The study is being conducted in compliance with the policies described in the study policies
- document, with the ethical principles that have their origin in the Declaration of Helsinki, with
- the protocol described herein, and with the standards of Good Clinical Practice (GCP).
- 184 Employing a cross-sectional registry component combined with the Natural History Study
- prospective longitudinal study design is advantageous because it reflects a systematic method of
- data collection. By doing so, this study addresses the need to evaluate disease progression while
- also accounting for prevalence and disease characteristics. This study design incorporates several
- strategies to minimize bias, detailed below, using considerations from "Rare Diseases: Natural
- History Studies for Drug Development: Guidance for Industry, Draft Guidance. 8 These are
- considered standard for treatment trials and will enhance the translation of the data from this
- 191 study to a treatment trial.
- 192 Establishing standardized testing procedures and specific required equipment for all
- investigators, leading to greater consistency and precision in the information collected.
- 194 Training and certification of study staff who will perform primary outcome procedures by a
- 195 Reading Center. The Reading Center will grade test results in a uniform manner independently
- 196 from study sites.
- 197 Use of standard, consistent definitions of pre-existing medical conditions, medications and
- treatments, and adverse events (AEs) across all clinical sites.
- A consistent schedule of follow-up visits for all participants with established visit time frames.
- 200 A coordinating center (CC) is responsible for monitoring the conduct of the study to ensure
- adherence to protocol.
- When feasible, data will be directly collected in electronic case report forms, which will be
- 203 considered the source data.

## Chapter 2: Registry Enrollment and Registry/Screening Visit

#### 2.1 Registry Recruitment and Enrollment

- 206 Registry participants will be recruited from approximately forty (40) clinical sites worldwide. All
- 207 eligible participants will be included without regard to gender, race, or ethnicity. The primary
- recruitment strategy will be patient referral from the site Investigator(s). However, recruitment
- materials may be made used upon IRB or Ethics Committee approval.
- The Executive Committee will review recruitment progress and feasibility at regular intervals.
- 211 Registry recruitment will continue until approximately 1,500 participants meet the final
- 212 **Registry Cohort Criteria** (see section 2.6), unless the Executive Committee terminates
- recruitment due to feasibility. The Executive Committee will monitor enrollment distributions
- 214 across genes, inheritance patterns, vision cohorts, and age cohorts with the planned caps as noted
- below. Enrollment in some genes, inheritance patterns, vision cohorts, or age cohorts may be
- 216 encouraged to ensure appropriate representation, and some caps may be adjusted if needed.

217218

219

220

221

222

223

224

225

226

227

228

229

230

231

232

233

234

235236

204

205

- A <u>maximum of 100</u> participants will be enrolled <u>within gene</u>.
- Recruitment will be tracked within the three (3) vision cohorts as defined below:
  - o A <u>maximum of 150</u> participants will be enrolled in Vision Cohort 3 (across genes).
  - Approximate target distribution of Vision Cohort 1 and 2 is 2:1 overall and within gene. This will be monitored and encouraged, but not required.
- A <u>maximum of 100</u> participants will be enrolled where Inheritance Pattern is Recessive and phase is unknown.
- Participants will <u>not</u> be counted as *enrolled into the Registry* until Genetic Screening Criteria have been confirmed (see section 2.5). This means that potentially more participants will complete the Registry/Screening Visit than are *enrolled into the Registry*. The number and reasons for screen failures will be tracked. It is possible that some participants will have completed the Registry/Screening Visit and will be awaiting genetic confirmation at the time the enrolled numbers reach the limits above. Therefore, the actual enrolled numbers may be larger. To limit over-enrollment, clinical sites will be notified as the recruitment limits are reached and efforts will be made to accurately predict numbers in the genetic screening queue.

#### 2.2 Cohort Definitions

#### **Vision Cohort Definitions**

| Vision Cohort 1 Approximately 900 participants | Criteria that must be met in the <b>better eye*</b> at the Registry/Screening Visit: o <b>visual acuity</b> ETDRS letter score of 54 or more (approximate Snellen equivalent 20/80 or better) <b>and visual field**</b> diameter 10 degrees or more in every meridian of the central field |
|---|---|
| Vision Cohort 2 Approximately 450 participants | Criteria that must be met in the <b>better eye*</b> at the Registry/Screening Visit: o <b>visual acuity</b> ETDRS letter score of 19-53 (approximate Snellen equivalent 20/100 to 20/400) OR |

| | o <b>visual acuity</b> ETDRS letter score of 54 or more (approximate Snellen equivalent 20/80 or better) <b>and visual field**</b> diameter less than 10 degrees in any meridian of the central field |
|---|---|
| <b>Vision Cohort 3</b> | Criteria that must be met in the <b>better eye*</b> at the Registry/Screening Visit: |
| Approximately | o visual acuity ETDRS letter score of 18 or less (approximate Snellen equivalent |
| 150 participants | 20/500 or worse) |
| *Better Eye | The <b>better eye</b> is defined as the eye with the better Registry/Screening Visit ETDRS visual acuity. However, if both eyes have the same visual acuity, which is defined as the same Snellen equivalent, then the determination will be made at the Investigator's discretion. In this scenario, the Investigator will consider the eye with better fixation or clearer ocular media to permit highest quality retinal imaging. |
| **Visual Field | The <b>visual field</b> (VF) is defined as the clinically determined <b>kinetic VF III4e</b> performed within the last 18 months prior to the Registry/Screening Visit or performed on the day of the Registry/Screening Visit. |

237238

#### Vision Cohort Grid

| | VF diameter ≥10° in | VF diameter <10° in |
|-----------------|---------------------|---------------------|
| | every meridian | any meridian |
| 20/80 or better | Vision Cohort 1 | Vision Cohort 2 |
| 20/100-20/400 | Vision Cohort 2 | Vision Cohort 2 |
| 20/500 or worse | Vision Cohort 3 | Vision Cohort 3 |

239240

#### **Younger Age Cohort Definition**

| Younger Age<br>Cohort | <ul> <li>Participants who are between the ages of ≥ 4 years and &lt; 8 years old will be designated as the Younger Age Cohort.</li> <li>Participants in this cohort will not be assigned a Vision Cohort.</li> <li>Registry/Screening Visit and Natural History Study Visits will have an abbreviated testing schedule.</li> </ul> |
|---|---|
|---|---|

#### 2.3 Registry Informed Consent and Authorization Procedures

There will be two separate consent processes for the two phases of the Uni-Rare study. There will be one (1) consent process for the Registry phase and one (1) for the NHS phase. The Registry consent process is as follows. Some sites outside the US may have alternative or additional Ethics Committee requirements, which will be followed as applicable, once reviewed and approved by the FFB Consortium.

247248

249

241

242

243244

245

246

Registry Consent Process for Age of Majority: For study participants who are the age of majority, e.g., at least eighteen (18) years of age in the US, the study will be discussed with the potential study participant by trained and delegated study staff. The potential

- study participant will be given the current, approved Registry Informed Consent Form (ICF) to read and will be given the opportunity to ask questions about the Registry. Potential study participants will be encouraged to discuss the study with family members and their personal physicians(s) before deciding whether to participate in the study. If the person wishes to be a participant, then the Registry ICF will be signed/dated and a signed/dated copy of the Registry ICF will be provided to the participant and another copy will be added to the participant's study record.
- Registry Consent Process for Minors: For potential participants who are minors, e.g., under eighteen (18) years of age in the US, a parent/legal guardian (referred to subsequently as "parent") will be provided with the Registry Informed Consent Form (ICF) to read and will be given the opportunity to ask questions about the Registry. If the parent agrees to participate, the Registry ICF will be signed/dated by the parent. The signed/dated Registry ICF will be provided to the parent and another copy will be added to the participant's study record. Participants who become age of majority, e.g., eighteen (18) years of age in the US, while in the Registry will need to re-consent with a Registry ICF (and authorization as described below), as applicable to the IRB or Ethics Committee requirements and as instructed by the FFB Consortium.

**Note:** Some Ethics Committees might require a separate Registry Assent for minors who are participating in the Registry, in addition to the Registry ICF signed by the parent/legal guardian. Such applicable requirements will be followed as instructed by the FFB Consortium.

Authorization for Use/Release of Personal Information: As part of the informed consent process, each participant and/or parent will be asked to sign/date an authorization for release of personal information (or other such document, e.g., HIPAA Authorization, GDPR Consent, LGPD Consent, etc.), as applicable to the IRB or Ethics Committee requirements. The trained and delegated study staff will review the study-specific information that will be collected and to whom that information will be disclosed. While speaking with the participant, questions will be answered about the details regarding authorization. If they wish to proceed, then they will receive a copy of the signed/dated authorization and another copy will be filed in the participant's study record.

#### > Other Consent Options:

- Short Form: If a participant or parent prefers that the study information be presented verbally/orally (e.g., they have significant visual impairments), a short form version of the Informed Consent Form, with the corresponding short form summary, may be used as approved by the IRB or Ethics Committee requirements and as instructed by the FFB Consortium.
  - Note: This process does require a witness. This process is not to be used as a substitute for presenting study information to the participant either due to written material not being translated in the native language of the participant/LAR or because a participant lacks the capacity to consent.
- <u>Remote Consent</u>: At the discretion of the site, as applicable to the IRB or Ethics Committee requirements, and with the approval of the FFB Consortium, some participants may complete the consent process remotely.

| 293<br>294 | <ul> <li>Note: This process typically requires additional documentation regarding<br/>the remote consent process (e.g., remote consent checklist).</li> </ul> | ng |
|---|---|---|
| | , | 440 |
| <ul><li>295</li><li>296</li></ul> | Completion of Consent Process and Enrollment: A participant is considered enrolled in initial screening when the Registry informed consent process has been completed and | |
| 290 | participant ID has been obtained on the study website. | а |
| 298 | 2.4 Registry/Screening Visit | |
| 299 | After the informed consent documents have been signed, the participant will be evaluated for | |
| 300 | study eligibility through the elicitation of a medical history and performance of ophthalmic tes | ts |
| 301 | as described below. The Registry/Screening Visit date will be documented as the date | |
| 302<br>303 | Registry/Screening procedures begin. All Registry/Screening Visit testing procedures must be completed within ninety (90) days of the Registry/Screening Visit date, unless specified below | ·• |
| 304 | 2.4.1 Registry Eligibility Criteria | |
| 305<br>306 | To be eligible to <i>enroll into the genetic screening phase</i> , a study participant must meet all the inclusion criteria and none of the exclusion criteria at the Registry/Screening Visit. | |
| 307 | 2.4.1.1 Participant Inclusion Criteria | |
| 308<br>309 | Participants must meet all the following inclusion criteria at the Registry/Screening Visit to be eligible to <i>enroll into the genetic screening phase</i> : | |
| 310 | 1. Willing to participate in the study and able to communicate consent during the consent | |
| 311 | process | |
| 312 | 2. Willing and able to complete all applicable <b>Registry/Screening Visit</b> assessments | |
| 313 | 3. Age $\geq$ 4 years | |
| 314 | 4. Must have a single gene on the RD Rare Gene List which meets one of the Genetic | |
| <ul><li>315</li><li>316</li></ul> | <b>Screening Criteria</b> below based on a genetic report* from a clinically certified lab (or from a research lab which has been approved by the study Genetics Committee): | |
| 317 | o Inheritance Pattern is Recessive <u>and</u> has at least 2 disease-causing variants which | ch |
| 318 | are homozygous or heterozygous in trans | |
| 319 | OR | |
| 320 | o Inheritance Pattern is Recessive <u>and</u> has 2 disease-causing variants with unknown | wn |
| 321 | phase <u>and</u> meets all the following additional informatic criteria that is consister | |
| 322 | with likely segregation in trans: | |
| 323 | 1. Investigator confirms genotype and phenotype are consistent with | |
| 324 | autosomal recessive inheritance | |
| 325 | 2. The 2 disease-causing variants have <b>not</b> been reported <i>in cis</i> in variant | |
| 326 | databases | 1 |
| 327 | 3. <u>No</u> additional potentially pathogenic variants were found on the gene (a the sequencing data for the gene were sufficiently robust to detect any | na |
| 328<br>329 | additional potentially pathogenic variants) | |
| 330 | 4. <b>No</b> potentially pathogenic variants were found in other common, likely | |
| 331 | candidate genes for the proposed condition | |
| 332 | OR | |

| 333<br>334<br>335 | <ul> <li>Inheritance Pattern is Dominant, X-linked, or Mitochondrial <u>and</u> has at least 1<br/>disease-causing variant</li> </ul> |
|---|---|
| 333 | Important Note: ➤ Genes Listed as Variable Mode of Inheritance on RD Rare Gene List ○ If the site is able to determine the inheritance pattern from the participant's genetic report*, the Genetic Screening Criteria above may be followed to determine eligibility based on the site determined inheritance pattern. ○ If the site is unable to determine the inheritance pattern from the participant's genetic report*, the site should use the most common inheritance pattern to follow the Genetic Screening Criteria above. The most common inheritance pattern will be provided to sites for each gene that is listed as having a variable mode of inheritance. ➤ If there are questions about interpretations of the genetic reports* prior to the genetic screening phase, the Genetics Committee (GC) and/or the Central Genetics Auditor (CGA) may be consulted. The Coordinating Center (CC) must be contacted first to determine the appropriate mechanism of consultation, consistent with regulatory and consent requirements. |
| 336<br>337 | *Genetic testing will not be performed in this study. A prior conclusive genetic test is what will be assessed for screening analysis. |
| 338 | 2.4.1.2 Ocular Inclusion Criteria |
| 339<br>340 | Both eyes must meet the following criteria at the Registry/Screening Visit to <i>enroll into the genetic screening phase</i> . |
| 341 | 1. Both eyes must have a clinical diagnosis of retinal dystrophy |
| 342<br>343 | 2. Both eyes must permit good quality photographic imaging (e.g., but not limited to, clear ocular media, adequate pupil dilation, stable fixation) |
| 344 | 2.4.1.3 Participant Exclusion Criteria |
| 345<br>346 | Participants must not meet any of the following exclusion criteria at the Registry/Screening Visit to be eligible to <i>enroll into the genetic screening phase</i> . |
| 347<br>348<br>349 | 1. History of more than 1 year of cumulative treatment, at any time, with an agent associated with pigmentary retinopathy including amiodarone, chloroquine, deferoxamine, hydroxychloroquine, pentosan polysulfate, tamoxifen, and deferoxamine |
| 350<br>351<br>352 | <b>Note:</b> Since this is an observational study, pregnant women will not be specifically excluded from participation. <b>However, minors that are pregnant shall be precluded from participation until they become the age of majority.</b> |
| 353 | 2.4.1.4 Ocular Exclusion Criteria |
| 354<br>355 | If either eye has any of the following ocular exclusion criteria at the Registry/Screening Visit, then the participant is not eligible to <i>enroll into the genetic screening phase</i> . |
| 356 | 1. Current vitreous hemorrhage |
| 357<br>358<br>359 | 2. Current complications of pathological myopia (for example, but not limited to, myopic maculopathy including atrophy, scar, choroidal neovascularization, schisis) that could inhibit ability to obtain good quality photographic imaging |

- 36. History of intraocular surgery (for example, but not limited to, cataract surgery, vitrectomy, penetrating keratoplasty, or LASIK) within 3 months of Registry/Screening Visit
  - **4.** Current or any history of confirmed diagnosis of glaucoma (for example, but not limited to, glaucomatous VF changes or nerve changes, or history of glaucoma filtering surgery)
  - 5. Current or any history of retinal vascular occlusion or proliferative diabetic retinopathy
  - **6.** History or current evidence of ocular disease that, in the opinion of the Investigator, may confound assessment of visual function (for example, but not limited to, tractional or rhegmatogenous retinal detachment, any vitreoretinal surgery, retinal vascular occlusion, proliferative diabetic retinopathy)
  - 7. The following medications and treatments are prohibited as they can affect progression of retinitis pigmentosa (RP). The participant must not have received the following treatments:
    - Any use of ocular stem cell or gene therapy
    - Any treatment with ocriplasmin

363

364

365

366

367

368

369

370

371

372

373374

375

376

377

378

379

380

381

382

383

390

391

394

395

396

398 399

400

- Treatment with Ozurdex (dexamethasone), Iluvien, or Yutiq (fluocinolone acetonide) intravitreal implant
- **8.** The following medications and treatments are excluded within the specified timeframe:
  - Treatment with an ophthalmic oligonucleotide within the last 9 months (last treatment date is less than 9 months prior to Registry/Screening Visit date)
  - ◆ Treatment with any other product within five times the expected half-life of the product (time from last treatment date to Registry/Screening Visit date is at least 5 times the half-life of the given product)

#### 2.4.2 Registry/Screening Visit Data Collection and Testing

- The following procedures will be performed at the Registry/Screening Visit. An overview of the
- equipment and certification requirements for all testing is in section 6.1. All Registry/Screening
- Visit testing procedures must be completed within ninety (90) days of the Registry/Screening
- Visit date, unless specified below. All ocular testing will be performed in each eye, right eye
- (OD) first and then left eye (OS). Screening procedures will last approximately two (2) hours.
- The testing procedures are detailed in the Uni-Rare Clinical Site Manual of Procedures.

#### All Registry/Screening Visit testing procedures are considered standard care.

- The following procedures will be performed and documented (including data collection and eligibility criteria checks) at the Registry/Screening Visit:
  - 1. Inclusion and exclusion criteria assessed
  - 2. Demographics (date of birth, sex, race, and ethnicity)
  - 3. Contact information (retained at the site and not entered on the study database)
- 4. Collection of MyRetinaTracker Registry ID (if participating and consented to provide)
  - 5. Medical history will be elicited from the study participant and extracted from available medical records, including patient-reported daily activities, pre-existing medical conditions, medications, and audiology history

| 402 | 7. Ophthalmic examination |
|---|---|
| Can be performed within ninety (90) days of the Registry/Screening historical measurement performed within the last six (6) months prior Registry/Screening Visit. | • Can be performed within ninety (90) days of the Registry/Screening Visit or a |
| | • |
| 406 | <ul> <li>Complete ophthalmic examination to include:</li> </ul> |
| 407 | Slit lamp biomicroscopy |
| 408 | <ul> <li>Indirect ophthalmoscopy</li> </ul> |
| 409 | 8. Visual acuity (including refraction, ETDRS, BRVT if needed, and LLVA if needed)* |
| 410<br>411 | • The VA letter score will determine whether LLVA or BRVT will be performed. The criteria are defined in the Uni-Rare Clinical Site Manual of Procedures. |
| 412 | 9. Intraocular Pressure (IOP) |
| 413 | • IOP measurements are to be taken prior to pupil dilation. |
| 414 | 10. Spectral Domain Optical Coherence Tomography (SD-OCT)* |
| 415 | ◆ Volume Scan |
| 416 | <ul> <li>Vertical and Horizontal Scan</li> </ul> |
| 417 | 11. Static Perimetry (SP)* |
| 418 | 12. Kinetic Visual Field III4e (Kinetic Perimetry [KP])* |
| 419 | • Vision Cohort 1 and 2: Historical measurement performed within the last |
| 420 | eighteen (18) months prior to the Registry/Screening Visit. If a historical |
| 421<br>422 | measurement is not available, then perform the Kinetic VF III4e during the Registry/Screening Visit. |
| 423 | • Vision Cohort 3: Collect the most recent historical measurement prior to the |
| Ų į | Registry/Screening Visit, if available. Kinetic VF III4e does not need to be |
| 425 | performed at screening if a historical measurement is not available. |
| 426 | 13. Determination of Vision Cohort (see section 2.2) |
| 427 | • If the participant's determined Vision Cohort is closed for enrollment, the remainder of procedures and testing are not required. Participant will be |
| 428<br>429 | discontinued as an <i>initial screen failure</i> . |
| 430 | <ul> <li>Participants in the Younger Age Cohort will not be assigned to a Vision Cohort.</li> </ul> |
| 431<br>432 | 14. Genetic screening assessment, including number and phase of mutations in the causal gene, history of consanguinity, and collection of the source genetic report(s) available at |
| 433 | the clinical site. |
| 434 | • This includes an assessment that the participant meets one of the <b>Genetic</b> |
| 435 | Screening Criteria. If the participant does not meet one of these criteria, then the |
| 436 | remainder of procedures and testing are not required. The participant will be |
| 437 | discontinued as an initial screen failure. |
| 438 | *This testing procedure will not be completed for participants in the Younger Age Cohort. |

6. Concomitant medications

401

| 439 | 2.4.3 Initial Screen Failures |
|---|---|
| 440<br>441<br>442<br>443 | Participants who do not meet criteria to continue as noted above will be discontinued as an <i>initial screen failure</i> . The Screening Visit Form will still be completed, entering "Not Done" for testing not finished. A Final Status Form will be completed, and the reason for screen failure will be noted. |
| 444 | 2.5 Genetic Screening Phase |
| 445<br>446<br>447<br>448 | Participants passing the initial screening and <i>enrolled into the genetic screening phase</i> will have their genetic lab reports submitted for Central Genetics Auditor (CGA) review. The schematic of study design at the beginning of the protocol summarizes the flow of the <b>Genetic Screening</b> Phase. Reference the Uni-Rare Clinical Site Manual of Procedures for detailed procedures. |
| 449<br>450<br>451<br>452<br>453 | All genetic reports will be uploaded to the FFB study website by the clinical site. These reports may be reviewed by the CC, associated clinical site, CGA, Genetics Committee, and Investigator(s) involved in the oversight of the study (which includes the study chair, Operations Committee, and Executive Committee). All genetic reports will be de-identified and redacted of all personal data prior to uploading on the FFB study website. |
| 454<br>455<br>456<br>457 | The CGA will review the genetic documentation provided by the clinical site to verify the genetic screening data entry and appropriate documentation of the <b>Genetic Screening Criteria</b> . Additional documentation, including relevant family history information, may be requested as needed to complete this verification process. |
| 458<br>459 | • If Genetic Screening Criteria are verified, then the participant will be considered enrolled into the Registry. |
| 460<br>461 | <ul> <li>If the final study cohort is not verified, then the participant will be a genetic screen<br/>failure.</li> </ul> |
| 462<br>463 | • <b>NOTE:</b> Genetic screen failures may include cases where CGA determines the following: |
| 464 | <ul> <li>More than one gene meets Genetic Screening Criteria</li> </ul> |
| 465<br>466<br>467 | • The actual inheritance pattern, according to CGA review, for the participant differs from the common designation on the <b>RD Rare Gene List</b> or identified by the site, and the associated <b>Genetic Screening Criteria</b> are no longer met |
| 468<br>469 | • Informatic criteria for Recessive with unknown phase is not confirmed to be consistent with segregation <i>in trans</i> |
| 470<br>471 | <ul> <li>Any of the inclusion/exclusion criteria under section 2.4.1 related to genetics<br/>are not met</li> </ul> |
| 472 | 2.5.1 Genetic Screen Failures |
| 473<br>474<br>475 | Participants who do not meet criteria to continue in the study will be discontinued as a <b>genetic screen failure</b> . A Final Status Form will be completed, and the reason for screen failure will be indicated. |

475

#### A Genetics Committee (GC) will review the genetic documentation of participants enrolled into 477 the Registry for interpretation and evaluation of whether the mutations in the affected gene are 478 causative of the disease (for example, pathogenic, likely pathogenic). Cases that are not 479

- confirmed as disease causing will remain in the study and will not be considered ineligible. 480
- 481 However, their data may be analyzed separately from those with pathogenic mutations.
- 482 2.6 Final Registry Cohort Criteria

476

2.5.2 Genetics Committee Review

- Participants who meet the Genetic Screening Criteria (section 2.4.1.1) and have those criteria 483
- confirmed by a CGA will be considered enrolled into the Registry. 484
## **Chapter 3: Registry Phase**

#### 3.1 Evaluation of Natural History Study (NHS) Target Gene Status

- Participants meeting criteria to *enroll into the Registry* (section 2.6) will be evaluated for NHS status.
  - ➤ If the participant's causal gene is designated as an **NHS Target Gene** at the time the CGA confirmation of Genetic Screening Criteria occurs, the participant will be considered *pending NHS* and will be asked to return to the clinical site for NHS Enrollment and Baseline Visit (procedures detailed in chapter 4).
  - ➤ If the participant's causal gene is <u>not</u> designated as an **NHS Target Gene** at the time the CGA confirmation of Genetic Screening Criteria occurs, the participant will remain active in the Registry Phase as follows:
    - Participants who are active in the Registry Phase will follow section 3.2 until the
      end of the Registry Phase of the study or until the participant's causal gene is
      designated as an NHS Target Gene.
    - When the causal gene is designated as an NHS Target Gene, the participant will be considered *pending NHS* and will be asked to return to the clinical site for NHS Enrollment and Baseline Visit (procedures detailed in chapter 4).

#### 3.2 Annual Phone Calls

485

486

489

490

491

492

493

494

495

496

497

498

499

500

501

502

508

509

510

The clinical site will call participants who are active in the Registry Phase annually according to the schedule below and will log the phone call on the study website. The purpose of the call is to maintain contact with the participant and update the participant on the status of the study, including any potential for their causal gene to become an NHS Target Gene or potential for interest in other studies.

#### **Schedule for Phone Calls**

| PHONE CALL<br>SCHEDULE | TARGET DATE* | TARGET<br>WINDOW* | ALLOWABLE<br>WINDOW* |
|---|---|---|---|
| 12-Month | 52 Weeks | ±8 Weeks | ± 26 Weeks |
| 24-Month | 104 Weeks | ± 8 Weeks | ± 26 Weeks |
| 36-Month | 156 Weeks | ± 8 Weeks | ± 26 Weeks |
| 48-Month | 208 Weeks | ± 8 Weeks | $\pm 26$ Weeks |

<sup>\*</sup>Timed from Registry/Screening Visit Date

#### 3.3 Completion of Registry Phase

- If a participant's causal gene has not been designated as an **NHS Target Gene** by the time of the
- 48-Month phone call, they will complete the Registry Phase and Uni-Rare study. The participant
- will be told on the 48-Month phone call that the annual study phone calls will discontinue and
- their study status will be complete. A Final Status Form will be completed.

## Chapter 4: Natural History Study Enrollment and Baseline Visit

#### 4.1 Natural History Study (NHS) Target Gene Selection

- The designation of **NHS Target Genes** will be made by the Executive Committee on an ongoing
- basis and may depend on funding resources as well as Registry enrollment numbers within gene.
- The Natural History Study sample size for each gene will depend on Registry enrollment. Since
- 520 the within-gene Registry limit is 100 participants, this will be the maximum sample size for NHS
- Target Genes. As noted in section 2.1, the actual enrolled numbers may be larger due to lag in
- genetic screening phase confirmation of participant meeting the final *Registry Cohort Criteria*.
- Within-gene sample size justification can be derived from the sample size estimates and
- statistical considerations in chapter 9.

#### 525 **4.2 NHS Enrollment**

- When a participant's causal gene is designated as an **NHS Target Gene**, the participant will be
- 527 considered *pending NHS* and will be asked to return to the clinical site for NHS Enrollment and
- 528 the Baseline Visit.

515

516

529

535

536

537

538

539

540

541

542

543

544

545

546

547

548

549

550

551

552

553

554

#### 4.2.1 NHS Informed Consent and Authorization Procedures

- There will be two separate consent process for the two phases of the Uni-Rare study. There will
- be one (1) consent process for the Registry phase and one (1) for the NHS phase. The NHS
- consent process is as follows. Some sites outside the US may have alternative or additional
- 533 Ethics Committee requirements which will be followed as applicable, once reviewed and
- approved by the FFB Consortium.
  - NHS Consent Process for Age of Majority: For study participants who are the age of majority, e.g., at least eighteen (18) years of age in the US, the study will be discussed with the potential study participant by trained and delegated study staff. The potential study participant will be given the current, approved NHS Informed Consent Form (ICF) to read and will be given the opportunity to ask questions about the NHS. Potential study participants will be encouraged to discuss the study with family members and their personal physicians(s) before deciding whether to participate in the study. If the person wishes to be a participant, then the NHS ICF will be signed/dated and a signed/dated copy of the NHS ICF will be provided to the participant and another copy will be added to the participant's study record.
  - NHS Consent Process for Minors: For potential participants who are minors, e.g., under eighteen (18) years of age in the US, a parent/legal guardian (referred to subsequently as "parent") will be provided with the NHS Informed Consent Form (ICF) to read and will be given the opportunity to ask questions about the NHS. If the parent agrees to participate, the NHS ICF will be signed/dated by the parent. The signed/dated NHS ICF will be provided to the parent and another copy will be added to the participant's study record. Participants who become age of majority, e.g., eighteen (18) years of age in the US, while in the NHS will need to re-consent with an NHS ICF (and authorization as described below), as applicable to the IRB or Ethics Committee requirements and as instructed by the FFB Consortium.

**Note:** Some Ethics Committees might require a separate NHS Assent for minors who are 555 participating in the Natural History Study, in addition to the NHS ICF signed by the 556 parent/legal guardian. Such applicable requirements will be followed as instructed by the 557 FFB Consortium. 558 Please reference section 2.3 for details regarding the Authorization for Use/Release of Personal 559 Information, Short Form Option, and Remote Consent Option. 560 561 4.2.2 NHS Eligibility Criteria To be eligible to *enroll into the NHS*, a study participant must meet the following criteria: 562 1. Enrolled into the Registry 563 a. Registry eligibility criteria (section 2.4.1) must be reviewed to confirm nothing 564 has changed and criteria are still met 565 b. Genetic Screening Criteria do not require a second review 566 2. Willing to participate in the Natural History Study and able to communicate consent 567 during the consent process 568 3. Willing and able to complete all Natural History Study visit assessments at each visit 569 over the forty-eight (48) month study period 570 4. Is <u>not</u> planning or expected to enter experimental treatment trial at any time during the 571 Natural History Study 572 5. Is not planning to receive any treatments or medications in either eye or systemically that 573 could affect progression of retinitis pigmentosa (RP), including the following: 574 • Any use of ocular stem cell or gene therapy 575 • Any treatment with ocriplasmin 576 • Treatment with Ozurdex (dexamethasone), Iluvien or Yutiq (fluocinolone acetonide) 577 intravitreal implant 578 A participant is considered *enrolled into the NHS* when the required NHS informed consent 579 document(s) have been signed, NHS eligibility criteria are confirmed, and an NHS Enrollment 580 Form is completed on the study website. This date is considered the NHS Enrollment Date. 581 Participants who do not meet criteria to continue as noted above will be discontinued as an NHS 582 screen failure. A Final Status Form will be completed, and the reason for screen failure will be 583 noted. 584 4.3 Baseline Visit Testing Procedures 585 The Baseline Visit must begin on or within seven (7) days of NHS Enrollment Date. The 586 Baseline Visit date will be documented as the date Baseline testing procedures begin. All 587 Baseline Visit testing procedures must be completed within thirty (30) days of the Baseline Visit 588 date, unless specified below. 589 The following procedures will be performed at the Baseline Visit. An overview of the equipment 590 591 and technician requirements for all testing is in section 6.1. All ocular testing will be performed

in each eye, right eye (OD) first and then left eye (OS). Baseline procedures will last

| 593<br>594 | | ely four (4) hours. The testing procedures are detailed in the <b>Uni-Rare Clinical Site Procedures</b> . |
|---|---|---|
| 595 | 4.3.1 Y | ounger Age Cohort |
| 596 | 1. | Medical updates to include: |
| 597 | | <ul> <li>New or changed adverse events (AEs)</li> </ul> |
| 598 | | New ocular procedures |
| 599 | | New or changed medications |
| 600 | 2. | Patient Reported Outcomes (PROs) |
| 601 | , | <ul> <li>ViSIO-ObsRO</li> </ul> |
| 602<br>603<br>604 | | • The PROs may be completed in person or remotely (phone or other remote methods) any time within six (6) months of the Baseline Visit (not required to be the same day as the rest of the Baseline Visit). |
| 605 | 3. | Complete ophthalmic examination to include: |
| 606 | | Slit lamp biomicroscopy |
| 607 | | Indirect ophthalmoscopy |
| 608<br>609<br>610<br>611 | | ◆ If the Baseline Visit date is within 3 months of the Registry/Screening Visit testing date and the ophthalmic examination was performed during the Registry/Screening Visit (i.e., not historical) − the ophthalmic examination testing procedure may be skipped. |
| 612 | 4. | Visual Acuity (including refraction, HOTV, BRVT if needed, LLVA if needed) |
| 613<br>614<br>615 | | • The visual acuity (VA) Snellen score will determine whether LLVA or BRVT will be performed. The criteria are defined in the Uni-Rare Clinical Site Manual of Procedures. |
| 616 | 5. | Intraocular Pressure (IOP) |
| 617 | | • IOP measurements are to be taken prior to pupil dilation. |
| 618<br>619 | | ◆ If the Baseline Visit date is within 3 months of the Registry/Screening Visit testing date – the IOP testing procedure may be skipped. |
| 620 | 6. | Color Vision |
| 621 | | • Desaturated (Lanthony D15) |
| 622 | 7. | Spectral Domain Optical Coherence Tomography (SD-OCT) |
| 623 | | ◆ Volume Scan |
| 624 | | Vertical and Horizontal Scan |
| 625<br>626<br>627 | | • If unable to perform OCT testing on the Heidelberg Spectralis, a site may use the handheld Bioptogen/Envisu to perform OCT testing for qualitative purposes with approval from the Coordinating Center. |
| 628 | 8. | Axial Length and Corneal Curvature Measurements |

| 629 | 9. Optos Color Photos* |
|---|---|
| 630 | 10. Optos Fundus Autofluorescence (FAF)* |
| 631 | 11. Full-field Electroretinogram (ffERG)* |
| 632 | 12. Full-field Stimulus Threshold (FST)* |
| 633<br>634<br>635 | <b>Note:</b> All testing procedures are to be <i>attempted</i> for participants in the Younger Age Cohort. If a child is unwilling to or unable to complete an examination, the procedure is to be skipped. |
| 636<br>637 | *If a site does not have the required equipment, participation in this test may be waived with approval from the Coordinating Center. |
| 638 | 4.3.2 Vision Cohorts 1 & 2 |
| 639 | 1. Medical updates to include: |
| 640 | <ul> <li>New or changed adverse events (AEs)</li> </ul> |
| 641 | <ul> <li>New ocular procedures</li> </ul> |
| 642 | <ul> <li>New or changed medications</li> </ul> |
| 643 | 2. Patient Reported Outcomes (PROs) |
| 644 | ◆ Adults (18+ years at Baseline): PROMIS®-29, MRDQ, ViSIO-PRO |
| 645 | • Adolescents (12-17 years at Baseline): LVP-FVQ II, ViSIO-PRO |
| 646 | • Children (8-11 years at Baseline): LVP-FVQ II, ViSIO-ObsRO |
| 647<br>648<br>649 | • The PROs may be completed in person or remotely (phone or other remote methods) any time within six (6) months of the Baseline Visit (not required to be the same day as the rest of the Baseline Visit). |
| 650 | 3. Complete ophthalmic examination to include: |
| 651 | Slit lamp biomicroscopy |
| 652 | ◆ Indirect ophthalmoscopy |
| 653<br>654<br>655<br>656 | ◆ If the Baseline Visit date is within 3 months of the Registry/Screening Visit testing date and the ophthalmic examination was performed during the Registry/Screening Visit (i.e., not historical) – the ophthalmic examination testing procedure may be skipped. |
| 657 | 4. Visual Acuity (including refraction, ETDRS, BRVT if needed, LLVA if needed) |
| 658<br>659<br>660 | <ul> <li>The visual acuity (VA) letter score will determine whether LLVA or BRVT will<br/>be performed. The criteria are defined in the Uni-Rare Clinical Site Manual of<br/>Procedures.</li> </ul> |
| 661<br>662 | ◆ If the Baseline Visit date is within 3 months of the Registry/Screening Visit<br>testing date – the VA testing procedure may be skipped. |
| 663 | 5. Intraocular Pressure (IOP) |
| 664 | • IOP measurements are to be taken prior to pupil dilation. |

| 665<br>666 | <ul> <li>If the Baseline Visit date is within 3 months of the Registry/Screening Visit<br/>testing date – the IOP testing procedure may be skipped.</li> </ul> |
|---|---|
| 667 | 6. Color Vision |
| 668 | <ul> <li>Desaturated (Lanthony D15)</li> </ul> |
| 669 | 7. Contrast Sensitivity |
| 670 | 8. Spectral Domain Optical Coherence Tomography (SD-OCT) |
| 671 | ◆ Volume Scan |
| 672 | Vertical and Horizontal Scan |
| 673<br>674 | <ul> <li>If the Baseline Visit date is within 3 months of the Registry/Screening Visit<br/>testing date – the SD-OCT testing procedure may be skipped.</li> </ul> |
| 675 | 9. Axial Length and Corneal Curvature Measurements |
| 676 | 10. Optos Color Photos* |
| 677 | 11. Optos Fundus Autofluorescence (FAF)* |
| 678 | 12. Full-field Electroretinogram (ffERG)* |
| 679 | 13. Full-field Stimulus Threshold (FST)* |
| 680 | 14. Static Perimetry (SP) |
| 681<br>682 | • Two (2) tests will be performed. The clinical site will compare the certified technician determined mean sensitivity from test one (1) versus test two (2). |
| 683<br>684<br>685 | (a) If the absolute value of the difference between the two tests is $\leq$ 2.4 dB, then the participant passes static perimetry reliability criteria. A third test is <u>not needed</u> . |
| 686 | <b>(b)</b> If the absolute value of the difference between the two tests is $> 2.4 \text{ dB}$ , |
| 687 | then the participant does not pass static perimetry reliability criteria. A |
| 688 | third test will be required. |
| 689 | • If the Baseline Visit date is within 3 months of the Registry/Screening Visit |
| 690 | testing date – the SP performed during the Registry/Screening Visit may be |
| 691 | considered the first test and does not need to be repeated. Only the second test |
| 692 | will need to be performed at the Baseline Visit; the need for a third test will be assessed using Test 1 from the Registry/Screening Visit and Test 2 from the |
| 693<br>694 | Baseline Visit. |
| 695 | 15. Fundus Guided Microperimetry (MP)* |
| 696 | • Two (2) tests will be performed. The clinical site will compare the certified |
| 697 | technician determined mean sensitivity from test one (1) versus test two (2). |
| 698 | (a) If the absolute value of the difference between the two tests divided by |
| 699 | the average between them is $\leq 50\%$ OR the absolute value of the |
| 700 | difference between the two tests is $\leq 0.5$ dB, then the participant passes |
| 701 | the microperimetry reliability criteria. A third test is not needed. |

| 702<br>703<br>704<br>705<br>706<br>707<br>708 | <ul> <li>(b) If the absolute value of the difference between the two tests divided by the average between them is &gt; 50% AND the absolute value of the difference between the two tests is &gt; 0.5 dB, then the participant does not pass microperimetry reliability criteria. A third test will be required.</li> <li>*If a site does not have the required equipment, participation in this test may be waived with approval from the Coordinating Center.</li> </ul> |
|---|---|
| 709 | 4.3.3 Vision Cohort 3 |
| 710 | 1. Medical updates to include |
| 711 | <ul> <li>New or changed adverse events (AEs)</li> </ul> |
| 712 | New ocular procedures |
| 713 | <ul> <li>New or changed medications</li> </ul> |
| | <u> </u> |
| 714 | 2. Patient Reported Outcomes (PROs) |
| 715<br>716 | <ul> <li>Adults (18+ years at Baseline): PROMIS®-29, MRDQ, ViSIO-PRO, ULV-VFQ-50</li> </ul> |
| 717 | <ul> <li>Adolescents (12-17 years at Baseline): LVP-FVQ II, ViSIO-PRO</li> </ul> |
| 718 | • Children (8-11 years at Baseline): LVP-FVQ II, ViSIO-ObsRO |
| 719 | • The PROs may be completed in person or remotely (phone or other remote |
| 720<br>721 | methods) any time within six (6) months of the Baseline Visit (not required to be the same day as the rest of the Baseline Visit). |
| 722 | 3. Complete ophthalmic examination to include: |
| 723 | Slit lamp biomicroscopy |
| 724 | <ul> <li>Indirect ophthalmoscopy</li> </ul> |
| 725 | • If the Baseline Visit date is within 3 months of the Registry/Screening Visit |
| 726 | testing date and the ophthalmic examination was performed during the |
| 727 | Registry/Screening Visit – the ophthalmic examination testing procedure may |
| 728 | be skipped. 4. Visual Assity (including refrection ETDDS DDVT if needed, LLVA if needed) |
| 729 | 4. Visual Acuity (including refraction, ETDRS, BRVT if needed, LLVA if needed) |
| 730<br>731 | ◆ The visual acuity (VA) letter score will determine whether LLVA or BRVT will be performed. The criteria are defined in the Uni-Rare Clinical Site Manual of |
| 732 | Procedures. |
| 733 | • If the Baseline Visit date is within 3 months of the Registry/Screening Visit |
| 734 | testing date – the VA testing procedure may be skipped. |
| 735 | 5. Intraocular Pressure (IOP) |
| 736 | <ul> <li>IOP measurements are to be taken prior to pupil dilation.</li> </ul> |
| 737<br>738 | ◆ If the Baseline Visit date is within 3 months of the Registry/Screening Visit<br>testing date – the IOP testing procedure may be skipped. |

| 739 | 6. Spectral Domain Optical Coherence Tomography (SD-OCT) |
|---|---|
| 740 | <ul> <li>Volume Scan</li> </ul> |
| 741 | Vertical and Horizontal Scan |
| 742<br>743 | <ul> <li>If the Baseline Visit date is within 3 months of the Registry/Screening Visit<br/>testing date – the SD-OCT testing procedure may be skipped</li> </ul> |
| 744 | 7. Axial Length and Corneal Curvature Measurements |
| 745 | 8. Optos Color Photos* |
| 746 | 9. Optos Fundus Autofluorescence (FAF)* |
| 747 | 10. Full-field Stimulus Threshold (FST)* |
| 748<br>749 | *If a site does not have the required equipment, participation in this test may be waived with approval from the Coordinating Center. |
| 750 | |
| 751 | |
| 752 | |

## **Chapter 5: Natural History Study Follow-up Visits**

#### 5.1 Follow-up Schedule

- 755 Follow-up Visits or phone calls will occur annually. Participants in the Younger Age Cohort
- 756 (YAC) and Vision Cohorts 1 and 2 will have annual in-person follow-up visits for four years
- after the Baseline Visit. Participants in Vision Cohort 3 will receive annual follow-up phone calls
- for three years after the Baseline Visit and will only return to the site for the last study visit (48-
- 759 Month Visit).

753

754

764

768

- The Baseline Visit date is considered study day zero (0) from which follow-up windows are
- timed. The Follow-up Visit date will be the date the Follow-up Visit testing procedures started.
- All Follow-up Visit testing procedures will be completed on the same date, other than the PROs
- as noted in Section 5.3 Follow-up Procedures.

#### **5.2 Target Timelines**

- Target dates and windows for each study Follow-up Visit for all cohorts are shown below. Dates and windows are timed from Baseline Visit date.
- 767 Schedule for Follow-up Visits or Phone Calls

| VISIT<br>SCHEDULE | VISIT TYPE | TARGET<br>DATE* | TARGET<br>WINDOW* | ALLOWABLE<br>WINDOW* |
|---|---|---|---|---|
| 12-Month | YAC + Vision Cohort 1 & 2:<br>In-person Visit | 52 Weeks | 4 3371 | ± 6 Weeks |
| 12-Monui | Vision Cohort 3:<br>Phone Call | 32 Weeks | ± 4 Weeks | |
| 24.36 4 | YAC + Vision Cohort 1 & 2:<br>In-person Visit | 104 Weeks | ± 4 Weeks | ± 6 Weeks |
| 24-Month | Vision Cohort 3:<br>Phone Call | 104 Weeks | | |
| 26 Manual | YAC + Vision Cohort 1 & 2:<br>In-person Visit | 156 W1 | ± 4 Weeks | ± 6 Weeks |
| 36-Month | Vision Cohort 3:<br>Phone Call | 156 Weeks | | |
| 48-Month | All Cohorts<br>In-person Visit | 208 Weeks | ± 4 Weeks | ± 6 Weeks |

<sup>\*</sup>Timed from Baseline Visit Date

- The goal is for all participants to complete all scheduled study visits. However, participants who
- (because of unforeseen circumstances) are unable or unwilling to return for all follow-up visits
- will be permitted to return for key visits only as an alternative to withdrawal from the study.
- Additional office visits may occur as needed.

#### 773 **5.3 Follow-up Visit Testing Procedures**

- The following procedures will be performed at the Follow-Up Visits, unless otherwise specified.
- An overview of the equipment and certification requirements for all testing is in section 6.1. All
- ocular testing will be performed in each eye, OD first and then OS. Follow-up Visit procedures
- will last approximately three (3) hours. The testing procedures are detailed in the Uni-Rare
- 778 Clinical Site Manual of Procedures.

779

780

781

786

787

788

789

790

791

792

793

794

795

796

797

799

803

804

805

806

#### 5.3.1 Younger Age Cohort

- 1. Medical updates to include:
- New or changed adverse events (AEs)
- 782 ◆ New ocular procedures
- New or changed medications 

  ◆ New or changed medications
- 784 2. Patient Reported Outcomes (PROs)
- 785 ♦ ViSIO-ObsRO
  - The PROs may be completed in person or remotely (phone or other remote methods) any time within the Allowable Window of the associated visit (not required to be the same day as the rest of the Follow-up Visit).
  - 3. Complete ophthalmic examination to include:
    - Slit lamp biomicroscopy
    - Indirect ophthalmoscopy
  - 4. Visual Acuity (including refraction, HOTV, BRVT if needed, LLVA if needed)
    - ◆ The visual acuity (VA) Snellen score will determine whether LLVA or BRVT will be performed. The criteria are defined in the Uni-Rare Clinical Site Manual of Procedures.
    - 5. Intraocular Pressure (IOP)
      - IOP measurements are to be taken prior to pupil dilation.
- 798 6. Color Vision
  - Desaturated (Lanthony D15)
- 7. Spectral Domain Optical Coherence Tomography (SD-OCT)
- 801 ◆ Volume Scan
- ♦ Vertical and Horizontal Scan
  - If unable to perform OCT testing on the Heidelberg Spectralis, a site may use the handheld Bioptogen/Envisu to perform OCT testing for qualitative purposes with approval from the Coordinating Center.
  - 8. Axial Length and Corneal Curvature Measurements
- 9. Optos Fundus Autofluorescence (FAF)\*

| 808 | 10. Full-field Electroretinogram (ffERG)* |
|---|---|
| 809 | <ul> <li>Complete at 48-Month Follow-up Visit Only</li> </ul> |
| 810 | 11. Full-field Stimulus Threshold (FST)* |
| 811 | 5.3.1.1 Age-Up Procedures |
| 812<br>813<br>814<br>815 | Participants in the Younger Age Cohort who turn 8 years old (age-up) during the NHS study period should attempt to have static perimetry, microperimetry, and contrast sensitivity testing performed at the next study visit after they turn 8 years old and at every subsequent visit, until the end of the study period. |
| 816 | 12. Static Perimetry (SP) |
| 817 | 13. Fundus Guided Microperimetry (MP)* |
| 818 | 14. Contrast Sensitivity |
| 819<br>820<br>821 | <b>Note:</b> All testing procedures are to be <i>attempted</i> for participants in the Younger Age Cohort. If a child is unwilling to or unable to complete an examination, the procedure is to be skipped. |
| 822<br>823 | *If a site does not have the required equipment, participation in this test may be waived with approval from the Coordinating Center. |
| 824 | 5.3.2 Vision Cohorts 1 & 2 |
| 825 | 1. Medical updates to include: |
| 826 | <ul> <li>New or changed adverse events (AEs)</li> </ul> |
| 827 | <ul> <li>New ocular procedures</li> </ul> |
| 828 | <ul> <li>New or changed medications</li> </ul> |
| 829 | 2. Patient Reported Outcomes (PROs) |
| 830 | <ul> <li>Complete at 24-Month and 48-Month Follow-up Visits Only</li> </ul> |
| 831 | • Adults (18+ years at Baseline): PROMIS®-29, MRDQ, ViSIO-PRO |
| 832 | <ul> <li>Adolescents (12-17 years at Baseline): LVP-FVQ II, ViSIO-PRO</li> </ul> |
| 833 | <ul> <li>Children (8-11 years at Baseline): LVP-FVQ II, ViSIO-ObsRO</li> </ul> |
| 834<br>835<br>836 | The PROs may be completed in person or remotely (phone or other remote<br>methods) any time within the Allowable Window of the associated visit (not<br>required to be the same day as the rest of the Follow-up Visit). |
| 837 | 3. Complete ophthalmic examination to include: |
| 838 | Slit lamp biomicroscopy |
| 839 | <ul> <li>Indirect ophthalmoscopy</li> </ul> |
| 840 | 4. Visual Acuity (including refraction, ETDRS, BRVT if needed, LLVA if needed) |

| 841<br>842<br>843 | <ul> <li>The visual acuity (VA) letter score will determine whether LLVA or BRVT will<br/>be performed. The criteria are defined in the Uni-Rare Clinical Site Manual of<br/>Procedures.</li> </ul> |
|---|---|
| 844 | 5. Intraocular Pressure (IOP) |
| 845 | • IOP measurements are to be taken prior to pupil dilation. |
| 846 | 6. Color Vision |
| 847 | <ul> <li>Desaturated (Lanthony D15)</li> </ul> |
| 848 | 7. Contrast Sensitivity |
| 849 | 8. Spectral Domain Optical Coherence Tomography (SD-OCT) |
| 850 | <ul> <li>Volume Scan</li> </ul> |
| 851 | <ul> <li>Vertical and Horizontal Scan</li> </ul> |
| 852 | 9. Axial Length and Corneal Curvature Measurements |
| 853<br>854 | <ul> <li>Only individuals who are under 18 years old at the Baseline Visit will continue to<br/>have measurements taken at every annual visit until study completion.</li> </ul> |
| 855 | 10. Optos Fundus Autofluorescence (FAF)* |
| 856 | 11. Full-field Electroretinogram (ffERG)* |
| 857 | <ul> <li>Complete at 48-Month Follow-up Visit Only</li> </ul> |
| 858 | 12. Full-field Stimulus Threshold (FST)* |
| 859 | 13. Static Perimetry (SP) |
| 860 | 14. Fundus Guided Microperimetry (MP)* |
| 861<br>862 | *If a site does not have the required equipment, participation in this test may be waived with approval from the Coordinating Center. |
| 863 | 5.3.3 Vision Cohort 3 |
| 864<br>865<br>866<br>867 | Phone contact will be scheduled at 12-, 24-, and 36-Month intervals. The purpose of the phone contact will be to keep the participants engaged in the study during the interim between the Baseline and 48-Month Follow-up Visits and to keep contact information updated. Changes in medications and AEs will also be collected. |
| 868 | The following will only be performed at 48-Month Visit: |
| 869 | 1. Medical updates to include |
| 870 | <ul> <li>New or changed adverse events (AEs)</li> </ul> |
| 871 | <ul> <li>New ocular procedures</li> </ul> |
| 872 | <ul> <li>New or changed medications</li> </ul> |
| 873 | 2. Patient Reported Outcomes (PROs) |
| 874<br>875 | <ul> <li>Adults (18+ years at Baseline): PROMIS®-29, MRDQ, ViSIO-PRO, ULV-VFO-50</li> </ul> |

| 876 | <ul> <li>Adolescents (12-17 years at Baseline): LVP-FVQ II, ViSIO-PRO</li> </ul> |
|---|---|
| 877 | • Children (8-11 years at Baseline): LVP-FVQ II, ViSIO-ObsRO |
| 878<br>879<br>880 | The PROs may be completed in person or remotely (phone or other remote<br>methods) any time within the Allowable Window of the associated visit (not<br>required to be the same day as the rest of the Follow-up Visit). |
| 881 | 3. Complete ophthalmic examination to include: |
| 882 | Slit lamp biomicroscopy |
| 883 | <ul> <li>Indirect ophthalmoscopy</li> </ul> |
| 884 | 4. Visual Acuity (including refraction, ETDRS, BRVT if needed, LLVA if needed) |
| 885<br>886<br>887 | <ul> <li>The visual acuity (VA) letter score will determine whether LLVA or BRVT will<br/>be performed. The criteria are defined in the Uni-Rare Clinical Site Manual of<br/>Procedures.</li> </ul> |
| 888 | 5. Intraocular Pressure (IOP) |
| 889 | <ul> <li>IOP measurements are to be taken prior to pupil dilation.</li> </ul> |
| 890 | 6. Spectral Domain Optical Coherence Tomography (SD-OCT) |
| 891 | <ul> <li>Volume Scan</li> </ul> |
| 892 | <ul> <li>Vertical and Horizontal Scan</li> </ul> |
| 893 | 7. Axial Length and Corneal Curvature Measurements |
| 894<br>895 | <ul> <li>Only individuals who were under 18 years old at the Baseline Visit will have<br/>measurements taken at 48M visit.</li> </ul> |
| 896 | 8. Optos Fundus Autofluorescence (FAF)* |
| 897 | 9. Full-field Stimulus Threshold (FST)* |
| 898<br>899 | *If a site does not have the required equipment, participation in this test may be waived with approval from the Coordinating Center. |
| 900 | 5.3.4 Unscheduled Visits |
| 901<br>902<br>903<br>904<br>905 | Testing procedures at unscheduled visits are at the Investigator's discretion. However, it is recommended that procedures performed during these visits follow the standard protocol for each procedure and be performed by certified personnel. Unscheduled visits will be recorded on the FFB Consortium study website. Study images taken during unscheduled visits do not require submission to the study website. |
| 906 | |

## **Chapter 6: Testing Procedures and Questionnaires**

## **6.1 Study Procedure Requirements**

907

908

909

910

911

The study procedure instructions are detailed in the **Uni-Rare Clinical Site Manual of Procedures**. An overview of the equipment and certification requirements for all testing are provided in the table below.

| Study Procedures | Description | Equipment<br>Required<br>(If applicable) | Site Personnel<br>Delegation |
|---|---|---|---|
| Investigator taking overall responsibility for a visit | Oversees that consent process was performed in accordance with IRB/EC requirements; signs off on all eCRFs for a participant, eCRF edits, and protocol deviations. | N/A | Certified investigator |
| Coordinator taking responsibility for the visit | Oversees the data entry aspect of the visit; addresses protocol queries and signs off on deviations. | N/A | Certified coordinator |
| Informed Consent Form<br>(ICF) Process | Explanation/review of study with the potential participant, including signature on the ICF. | N/A | Certified investigator or coordinator as permitted by the IRB/EC |
| Signature of Informed<br>Consent Form | The participant and/or LAR sign the ICF. The person obtaining the ICF will also sign. | N/A | Certified investigator or coordinator as permitted by the IRB/EC |
| Data entry on study<br>website | Data collected from the study participant will be directly entered on the FFB Study Website (strongly encouraged) or written on the paper CRF and transcribed on the FFB Study Website within seven (7) days. | Computer and internet connection | Certified coordinator or certified investigator with additional study website certification |
| Collect information regarding medical history, demographics, adverse events, medications | Sites will collect medical history, demographic information, Aes, and medications from the participant during each visit. This information can be confirmed by requesting medical records if needed. | N/A | Certified investigator or coordinator |
| Patient Reported Outcome (PRO) | There are six (6) questionnaires depending on age and Vision Cohort (details in section 6.2). | Study will provide | Certified investigator or coordinator |
| Ocular Exam | Including slit lamp biomicroscopy and indirect ophthalmoscopy | Any equipment is acceptable | Certified investigator |
| Intraocular Pressure<br>(IOP) | Measurement of the fluid pressure inside the eye | Any equipment is acceptable | Clinical site personnel performing this test does not require a study specific certification. However, they must be trained and delegated by the PI per the SSDL. |

| Study Procedures | Description | Equipment<br>Required<br>(If applicable) | Site Personnel<br>Delegation |
|---|---|---|---|
| Visual Acuity –<br>Refraction | Refraction is done as a routine part of an eye exam to achieve best corrected visual acuity measures. | N/A | Clinical site personnel certified for refraction |
| Visual Acuity – ETDRS | Traditional measure of central visual function that represents foveal cone function. | EVA system or<br>ETDRS charts | Clinical site personnel certified for VA (including ETDRS) |
| Visual Acuity – LLVA | Measures vision function in low luminance conditions | EVA system or<br>ETDRS charts<br>2.0 neutral<br>density filter to<br>be provided by<br>study | Clinical site personnel certified for VA (including LLVA) |
| Visual Acuity – BRVT | A three-level hierarchy for visual acuity testing better suited for low vision participants | BRVT charts<br>provided by<br>study | Clinical site personnel certified for BRVT |
| Visual Acuity – HOTV | Pediatric measure of central visual function that represents foveal cone function. | HOTV chart and<br>lap card<br>provided by<br>study | Clinical site personnel certified for VA (including HOTV) |
| Color Vision | Measures the type and severity of color blindness | Lanthony D15<br>provided by<br>study | Clinical site personnel performing this test does not require a study specific certification. However, they must be trained and delegated by the PI per the SSDL. |
| Contrast Sensitivity | Measure ability to distinguish between increments of light versus dark | CSV-1000E<br>provided by<br>study | Clinical site personnel performing this test does not require a study specific certification. However, they must be trained and delegated by the PI per the SSDL. |
| Spectral Domain Optical<br>Coherence Tomography<br>(SD-OCT) – Volume Scan | Scans provide objective, non-<br>invasive measures of retinal<br>structure | Heidelberg<br>Spectralis** | Clinical site personnel certified for SD-OCT |
| Spectral Domain Optical<br>Coherence Tomography<br>(SD-OCT) – Vertical and<br>Horizontal Scan | Scans provide objective, non-<br>invasive measures of retinal<br>structure | Heidelberg<br>Spectralis** | Clinical site personnel certified for SD-OCT and vertical and horizontal scan |
| Axial Length and Corneal<br>Curvature | Axial length measures the distance between the anterior and posterior poles of the eye. Corneal curvature determines the power of the cornea. | Any equipment is acceptable | Clinical site personnel performing this test does not require a study specific certification. However, they must be trained and delegated by the PI per the SSDL. |

| Study Procedures | Description | Equipment<br>Required<br>(If applicable) | Site Personnel<br>Delegation |
|---|---|---|---|
| <b>Optos Color Photos</b> | Images provide objective, non-<br>invasive visualization of the<br>photoreceptor layer and RPE | Optos* | Clinical site personnel certified for Optos Color photos |
| Optos Fundus<br>Autofluorescence (FAF) | Images provide objective, non-<br>invasive map of lipofuscin in RPE | Optos* | Clinical site personnel certified for Optos FAF |
| Full-field Electroretinogram (ffERG) | Measures rod- and cone-mediated parts of the visual field | Diagnosys<br>Espion* | Clinical site personnel certified for ffERG |
| Full-field Stimulus<br>Threshold (FST) | Measures rod- and cone-mediated parts of the visual field | Diagnosys<br>Espion* | Clinical site personnel performing this test does not require a study specific certification. However, they must be trained and delegated by the PI per the SSDL. |
| Static Perimetry (SP) | Measures sensitivity thresholds at specified test locations | Octopus 900 Pro<br>(GATE<br>Protocol) | Clinical site personnel certified for SP |
| Fundus guided<br>microperimetry (MP) | Measures sensitivity thresholds at specified test locations | MAIA* | Clinical site personnel certified for MP |
| Kinetic Perimetry (KP) | Measures sensitivity thresholds at specified test locations | Any equipment is acceptable | (Historical) Does not need<br>to be performed by study<br>certified personnel or<br>recorded in the SSDL |

- \*If site does not have required equipment, participation in this test may be waived with
- 913 approval from the Coordinating Center
- \*\*If Younger Age Cohort participant is unable to perform OCT testing on the Heidelberg
- Spectralis, a site may use the handheld Bioptogen/Envisu to perform OCT testing for qualitative
- purposes with approval from the Coordinating Center.

#### 917 **6.2 Questionnaires**

- The following questionnaires will be administered in the study by a certified investigator or
- coordinator. Each questionnaire takes about 15 minutes to administer.

| Questionnaire | Type | Description | Vision<br>Cohort | Age at<br>Baseline |
|---|---|---|---|---|
| Michigan Retinal<br>Degeneration<br>Questionnaire<br>(MRDQ) | Vision<br>Function | The MRDQ is a psychometrically validated patient-reported outcome measure for inherited retinal degenerations questionnaire which consists of fifty-nine (59) questions measuring seven (7) unidimensional domains: central vision, color vision, contrast sensitivity, scotopic function, photopic peripheral vision, mesopic peripheral vision, and photosensitivity. | All | Adults<br>≥18 years |

| PROMIS-29®<br>(Patient-Reported<br>Outcomes<br>Measurement<br>Information<br>System®) | Global<br>Physical,<br>Mental,<br>and Social<br>Health | The PROMIS®-29 contains items from seven PROMIS domains: depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities. The seven domains cover the most relevant areas of self-reported health for most people with chronic illness. There is also one 11-point rating scale for pain intensity. | All | Adults<br>≥18 years |
|---|---|---|---|---|
| Visual Symptom<br>and Impact<br>Outcomes Patient<br>Reported Outcome<br>(ViSIO-PRO) | Vision<br>Function<br>and<br>HRQoL | The ViSIO-PRO instrument is designed to assess visual function symptoms, impacts on functional vision, and impacts on wider health-related quality of life (HRQoL). It has been designed for completion by adolescents (12-17) and adults (18 +) with retinitis pigmentosa (RP). | All | Adolescents<br>(12-17 years)<br>& Adults<br>(≥18 years) |
| Visual Symptom<br>and Impact<br>Outcomes Observer<br>Reported Outcome<br>(ViSIO-ObsRO) | Vision<br>Function<br>and<br>HRQoL | The ViSIO-ObsRO instrument is designed to assess visual function symptoms, impacts on functional vision, and impacts on wider health-related quality of life (HRQoL). It has been designed for completion by parents/caregivers of children with retinitis pigmentosa (RP) aged 3-11 years. | All | Children<br>4-11 years |
| L. V. Prasad-<br>Functional Vision<br>Questionnaire<br>(LVP-FVQ II) | Vision<br>Function | The LVP-FVQ-II questionnaire consists of 23 questions. The questionnaire is used to assess self-reported difficulties in performing daily tasks in children with visual impairment. | All | Adolescents<br>(12-17 years)<br>& Children<br>(8-11 years) |
| Ultra-Low Vision<br>Visual Functioning<br>Questionnaire<br>(ULV-VFQ-50) | Vision<br>Function | The ULV-VFQ-50 psychometrically evaluates a visual functioning questionnaire (VFQ) in an ultralow vision (ULV) population | Vision<br>Cohort<br>3 | Adults<br>≥18 years |

| 921<br>922 | Chapter 7: Unanticipated Problem and Adverse Event Reporting |
|---|---|
| 922 | Auverse Event Reporting |
| 923 | 7.1 Unanticipated Problems |
| 924<br>925<br>926<br>927<br>928 | Site investigators will promptly report all unanticipated problems meeting the criteria below on an electronic case report form (eCRF). Sites overseen by the JCHR IRB must report Unanticipated Problems to the IRB within seven (7) calendar days of recognition. For this protocol, an unanticipated problem is an incident, experience, or outcome that meets all the following criteria: |
| 929<br>930<br>931<br>932 | <ul> <li>Unexpected (in terms of nature, severity, or frequency) given (a) the research<br/>procedures that are described in the protocol related documents, such as the IRB-<br/>approved research protocol and informed consent document; and (b) the<br/>characteristics of the subject population being studied.</li> </ul> |
| 933<br>934<br>935 | • Related or possibly related to participation in the research (possibly related means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research). |
| 936<br>937<br>938 | <ul> <li>Suggests that the research places participants or others at a greater risk of harm than was previously known or recognized (including physical, psychological, economic, or social harm).</li> </ul> |
| 939<br>940<br>941 | The Coordinating Center also will report to the IRB all unanticipated problems not directly involving a specific site such as unanticipated problems that occur at the Coordinating Center or at another participating entity such as a laboratory. |
| 942<br>943<br>944<br>945<br>946 | These instances must be reported to the JCHR IRB within seven (7) calendar days of recognition. The Director of the Human Research Protection Program (HRPP) will report to the appropriate regulatory authorities if the IRB determines that the event indeed meets the criteria of an Unanticipated Problem that requires further reporting to fulfill the reporting obligations of the HRPP. |
| 947 | 7.2 Adverse Events |
| 948<br>949 | The following section on adverse events applies to the Natural History Study phase of the study. |
| 950 | 7.2.1 Definitions |
| 951<br>952 | <b>Adverse Event (AE):</b> Any untoward medical occurrence (including laboratory findings) associated with study procedures whether the event is considered related. |
| 953<br>954 | <b>Serious Adverse Event (SAE):</b> Any untoward medical occurrence that results in any of the following outcomes: |
| 955 | • Death. |
| 956<br>957<br>958 | ◆ A life-threatening adverse event: (a non-life-threatening event which, had it been more severe, might have become life-threatening, is not necessarily considered a serious adverse event). |

- Inpatient hospitalization or prolongation of existing hospitalization.
  - A persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions.
    - A congenital anomaly or birth defect.
- An important medical event that may not result in death, be life-threatening, or require
- hospitalization may be considered serious when, based upon appropriate medical judgment, they
- may jeopardize the patient or subject and may require medical and surgical intervention to
- prevent one of the outcomes listed in this definition.
- Note: As this is a Natural History Study, the Investigator(s) will make the categorical
- determinations of Adverse Events, as described above, and will report each determination to the
- 969 Coordinating Center, as per data collection.

#### 7.2.2 Reportable Adverse Events

- For this protocol, a reportable adverse event includes all events meeting the definition of an
- 972 adverse event.

960

961

962

970

981

- All reportable Adverse Events whether volunteered by the participant, discovered by study
- personnel during questioning, or detected through ophthalmological examination, laboratory test,
- or other means will be reported on an adverse event form online.
- The purpose of AE collection for the Uni-Rare study will be to provide historical controls for
- 977 future clinical trials. As a no greater than minimal risk study, AEs do not require any specific
- 978 reporting to regulatory or oversight bodies. However, each Principal Investigator (PI) is
- 979 responsible for abiding by any other reporting requirements specific to their IRB or equivalent
- 980 ethics oversight committee.

#### 7.2.3 Relationship of Adverse Event to Study Procedure

- The study Investigator(s) will assess the relationship of any adverse event to be related or
- unrelated to a study procedure by determining if there is a reasonable possibility that the adverse
- event may have been caused by the study procedure.
- To ensure consistency of adverse event causality assessments, the Investigator(s) should apply
- the following general guideline when determining whether an adverse event is related:
- 987 **Yes**
- There is a plausible temporal relationship between the onset of the adverse event and the study
- procedure, and the adverse event cannot be readily explained by the participant's clinical state,
- intercurrent illness, or concomitant therapies; and/or the adverse event follows a known pattern
- of response to the study procedure; and/or the adverse event abates or resolves upon
- 992 discontinuation of the study procedure.
- 993 **No**
- Evidence exists that the adverse event has an etiology other than the study procedure (for
- example, preexisting medical condition, underlying disease, intercurrent illness, or concomitant
- medication); and/or the adverse event has no plausible temporal relationship to study procedure.

| 997 | 7.2.4 \$ | Severity (Intensity) of Adverse Event |
|---|---|---|
| 998<br>999<br>1000 | adverse ev | assessment is a clinical determination of the intensity of an event. Thus, a severe vent is not necessarily serious. For example, itching for several days may be rated as t may not be clinically serious. |
| 1001<br>1002 | | ity (intensity) of an adverse event will be rated on a three-point scale: (1) mild, (2) or (3) severe. |
| 1003<br>1004 | 1. | <b>MILD:</b> Usually transient, requires no special treatment, and does not interfere with the participant's daily activities. |
| 1005<br>1006<br>1007 | 2. | <b>MODERATE:</b> Usually causes a low level of inconvenience, discomfort or concern to the participant and may interfere with daily activities but is usually ameliorated by simple therapeutic measures and participant is able to continue in study. |
| 1008<br>1009 | 3. | <b>SEVERE:</b> Interrupts a participant's usual daily activities and causes severe discomfort. |
| 1010 | 7.2.5 1 | Expectedness |
| 1011<br>1012 | As this is assessed. | a Natural History Study, the expectedness for a serious adverse event will not be |
| 1013 | 7.2.6 | Coding of Adverse Events |
| 1014<br>1015 | | vents will be coded using the Medical Dictionary for Regulatory Activities 1). To facilitate coding, the site will enter a preliminary MedDRA code |
| 1016 | 7.2.7 | Outcome of Adverse Event |
| 1017 | The outco | me of each reportable adverse event will be classified by the Investigator(s) as follows: |
| 1018<br>1019 | 1. | <b>RECOVERED/RESOLVED (COMPLETE RECOVERY)</b> – The participant recovered from the AE/SAE without sequelae. Record the AE/SAE stop date. |
| 1020<br>1021<br>1022 | 2. | <b>RECOVERED/RESOLVED WITH SEQUELAE</b> – AE/SAE where the subject recuperated but retained pathological conditions resulting from the prior disease or injury. Record the AE/SAE stop date. |
| 1023<br>1024<br>1025<br>1026 | 3. | <b>FATAL</b> – A fatal outcome is defined as the SAE that resulted in death. Only the event that was the cause of death should be reported as fatal. AEs/SAEs that were ongoing at the time of death; however, were not the cause of death, will be recorded as "resolved" at the time of death. |
| 1027<br>1028 | 4. | <b>ONGOING NOT RECOVERED/NOT RESOLVED</b> – An ongoing AE/SAE is defined as an ongoing event with an undetermined outcome. |
| 1029<br>1030 | | • An ongoing outcome will require follow-up by the site in order to determine the final outcome of the AE/SAE. |
| 1031<br>1032<br>1033 | | • The outcome of an ongoing event at the time of death that was not the cause of death, will be updated and recorded as "resolved" with the date of death recorded as the stop date. |

| 1034<br>1035 | 5. <b>ONGOING (MEDICALLY STABLE)</b> – AE/SAE is ongoing, but medically stable. For example, a chronic condition where no further change is expected. |
|---|---|
| 1036<br>1037<br>1038<br>1039<br>1040 | If any reported adverse events are ongoing when a participant completes the study (or withdraws), they will be followed until they are either resolved, or have no prospect of improvement or change, even after the participant has completed all applicable study visits/contacts. For all other adverse events, data collection will end at the time the participant completes the study. |
| 1041<br>1042 | <b>Note:</b> Participants should continue to receive appropriate medical care for an adverse event after their participation in the study ends. |
| 1043<br>1044 | If a participant is lost to follow up and participant outcome cannot be determined, outcome classification will be the last known outcome. |
| 1045 | 7.3 Timing of Event Reporting |
| 1046<br>1047 | Investigator(s) are responsible for reporting Adverse Events on the electronic case report form (eCRF) through the study website in a timely manner. |
| 1048<br>1049<br>1050<br>1051<br>1052 | Each Principal Investigator (PI) is responsible for reporting serious study-related adverse events and abiding by any other reporting requirements specific to his/her Institutional Review Board (IRB) or Ethics Committee (EC). Where the JCHR IRB is the overseeing IRB, sites must report all serious, related adverse events regardless of whether they are expected/anticipated and regardless of whether they are fatal or life-threatening within seven (7) calendar days. |
| 1053 | |

| 1054 | <b>Chapter 8: Miscellaneous Considerations</b> |
|---|---|
| 1055 | 8.1 New or Ongoing Medical Conditions and Medications |
| 1056 | 8.1.1 Pre-Existing Conditions |
| 1057<br>1058<br>1059 | Any medical condition that is either present at screening, a chronic disease, or a prior condition that could impact the participant's health during the study (for example, prior myocardial infarction or stroke). |
| 1060 | 8.1.2 Medications |
| 1061<br>1062<br>1063<br>1064 | All medication for the treatment of chronic pre-existing conditions, medical conditions, and/or adverse events that the participant is currently taking at screening and during the study should be recorded. Certain nutraceuticals and preventative treatments that are of interest to the study should also should be recorded. |
| 1065 | 8.1.3 Medical Conditions During the Natural History Study |
| 1066<br>1067<br>1068<br>1069<br>1070 | In addition to conditions meeting the reporting requirements for an adverse event or as described above, the following medical conditions should also be reported: (1) new diagnosis of a chronic disease (for example, not present at the time of enrollment), and (2) any medical condition that could affect the participant's ability to carry out any aspect of the protocol or could affect an outcome assessment. These will be reported as adverse events. See chapter 7 for more detail. |
| 1071 | 8.2 Prohibited Medications, Treatments, and Procedures During the Natural History Study |
| 1072 | 8.2.1 Prohibited Medications and Treatment for Retinal Degeneration |
| 1073<br>1074<br>1075<br>1076<br>1077 | Participants who are <i>enrolled into the NHS</i> should not administer IRD treatments during the study. This includes enrolling into an experimental treatment trial of underlying conditions related to the causal gene during the 4-year study duration. However, if the participants enroll in a treatment trial the Executive Committee will be consulted and will determine if the participant will continue in the study. |
| 1078<br>1079<br>1080<br>1081<br>1082<br>1083<br>1084 | Examples of prohibited medications and treatments include, but are not limited to the following: • use of ocular stem cell or gene therapy • ocriplasmin • ophthalmic oligonucleotide • Ozurdex (dexamethasone) • Iluvien • Yutiq (fluocinolone acetonide) intravitreal implant |
| 1085 | 8.2.2 Intraocular Surgical Procedures |
| 1086<br>1087<br>1088<br>1089<br>1090 | Participants <i>enrolled into the NHS</i> , who have intraocular surgery during the study, will have follow-up visits timed either before the surgery date or at least three (3) months after the surgery date, to minimize the impact on the natural history outcome measures. Clinical sites will make reasonable efforts to schedule the participant's follow-up visit as close to the visit target window as possible. |

| 091 | 8.2.3 Treatment for Cystoid Macular Edema (CME) |
|---|---|
| 092 | Participants <i>enrolled into the NHS</i> , who need to receive treatment for CME during the study, may do so without affecting their participation in the study. |
| .094 | 8.3 Pregnancy Reporting |
| 095<br>096<br>097<br>098<br>099<br>100 | If a pregnancy occurs, the participant will remain in the study. The occurrence of pregnancy will be reported to the Coordinating Center within seven (7) days of the site's discovery of the pregnancy (including at screening) and the Confirmed Pregnancy Notification Worksheet will be completed within seven (7) calendar days. Sites will collect concomitant medications throughout the pregnancy. If an Adverse Event occurs because of the pregnancy, then the site will record the Adverse Event on the Adverse Event form. |
| 101 | 8.4 Participant Compensation |
| 102 | Participant compensation will be specified in the informed consent form. |
| 103 | 8.5 Participant Withdrawal |
| 104 | Participation in the study is voluntary, and a participant may withdraw at any time. For participants who withdraw, their data will be used up until the time of withdrawal. |
| 106 | 8.6 Confidentiality |
| 107<br>108<br>109 | For security and confidentiality purposes, participants will be assigned an identifier that will be used instead of their name. Protected health information (PHI) gathered for this study will be shared with the coordinating center, the Jaeb Center for Health Research in Tampa, FL. Deidentified participant information may also be provided to research sites involved in the study |

## **Chapter 9: Statistical Considerations**

The approach to sample size (N) and statistical analyses are summarized below.

#### 9.1 Sample Size Approach

1111

1113

1116

1126

1127

1132

1133

1134

1135

1136

1137

1138

1139

1140

1141

1142

The following is a framework for evaluating and justifying within-gene sample size for any gene in the Uni-Rare Study.

#### 9.1.1 General Considerations

Both eyes of a participant will be assessed for the main ocular measures of interest. Thus, if there 1117 are N participants, 2N eyes will be available for analysis. However, outcome measures from two 1118 (2) eyes of a person are typically strongly correlated ( $r \ge 0.5$ ). The contribution of information 1119 from the two (2) eyes in this case is (2/(1+r)) instead of two (2). Values for the multiplier to the 1120 number of participants to obtain an effective sample size are given below in **Table 9-1**. The 1121 correlation between eyes (inter-eye correlation) for each outcome measure is not known. We 1122 assume an inter-eye correlation of 0.8 throughout all sample size calculations throughout section 1123 1.1. This assumption is conservative in that it requires a higher number of participants than lower 1124 plausible values of r. 1125

#### Table 9-1. Multiplier to Obtain Effective N Based on Inter-Eye Correlation

| r | 0.0 | 0.1 | 0.2 | 0.3 | 0.4 | 0.5 | 0.6 | 0.7 | 0.8 | 0.9 | 1.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Multiplier for<br>Effective N | 2.00 | 1.82 | 1.67 | 1.54 | 1.43 | 1.33 | 1.25 | 1.18 | 1.11 | 1.05 | 1.00 |

#### 9.1.2 Registry Sample Size Considerations

As noted in section 2.1, the Registry recruitment will remain open until a total of 1,500 participants meeting *Registry Cohort Criteria* are enrolled, with **a maximum of 100** participants enrolled within any gene. The following Registry sample size considerations focus on Registry Objective 2 (see section 1.3).

#### Registry Objective 2 (Cross-Sectional Phenotype Characterization)

- **Registry Objective 2** is to characterize cross-sectional retinal dystrophy associated with disease-causing genetic variants using functional and structural measures, **within gene**.
- For a given gene, the potential sample size for the gene will impact the precision around the point estimates for the key measures of interest.
- ➤ Table 9-2, 9-3, and 9-4 provide the half-width of the 95% confidence interval (CI) around the estimated cross-sectional mean value, for three key measures of interest (visual acuity, OCT EZ area, and SP V<sub>tot</sub>, respectively) under different possible sample sizes and standard deviations (SD) of the distribution of the cross-sectional measure. The larger the SD and/or the smaller the sample size, the wider the CI, meaning the range of possible true values grows.

# Table 9-2. Half-Width of 95% Confidence Intervals Around the Estimated Mean Cross-Sectional Visual Acuity

| | | Sample Size | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | (effective sample size after adjusting for inter-eye correlation $r=0.8$ ) | | | | | | | | |
| | N=10 | N=20 | N=30 | N=40 | N=50 | N=60 | N=70 | N=80 | N=90 | N=100 |
| | (11) | (22) | (33) | (44) | (56) | (67) | (78) | (89) | (100) | (111) |
| SD=5 | 3.4 | 2.2 | 1.8 | 1.5 | 1.3 | 1.2 | 1.1 | 1.1 | 1.0 | 0.9 |
| SD=10 | 6.7 | 4.4 | 3.5 | 3.0 | 2.7 | 2.4 | 2.3 | 2.1 | 2.0 | 1.9 |
| SD=15 | 10.1 | 6.7 | 5.3 | 4.6 | 4.0 | 3.7 | 3.4 | 3.2 | 3.0 | 2.8 |
| SD=20 | 13.4 | 8.9 | 7.1 | 6.1 | 5.4 | 4.9 | 4.5 | 4.2 | 4.0 | 3.8 |

1145 Units = letter score

1143 1144

#### 1146 Table 9-3. Half-Width of 95% Confidence Intervals Around the Estimated Mean Cross-

#### 1147 Sectional OCT Ellipsoid Zone Area

| | | Sample Size | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | (effective sample size after adjusting for inter-eye correlation $r$ =0.8) | | | | | | | | |
| | N=10 | N=20 | N=30 | N=40 | N=50 | N=60 | N=70 | N=80 | N=90 | N=100 |
| | (11) | (22) | (33) | (44) | (56) | (67) | (78) | (89) | (100) | (111) |
| SD=2 | 1.3 | 0.9 | 0.7 | 0.6 | 0.5 | 0.5 | 0.5 | 0.4 | 0.4 | 0.4 |
| SD=5 | 3.4 | 2.2 | 1.8 | 1.5 | 1.3 | 1.2 | 1.1 | 1.1 | 1.0 | 0.9 |
| SD=8 | 5.4 | 3.5 | 2.8 | 2.4 | 2.1 | 2.0 | 1.8 | 1.7 | 1.6 | 1.5 |
| SD=10 | 6.7 | 4.4 | 3.5 | 3.0 | 2.7 | 2.4 | 2.3 | 2.1 | 2.0 | 1.9 |

1148 Units =  $mm^2$ 

#### 1149 Table 9-4. Half-Width of 95% Confidence Intervals Around the Estimated Mean Cross-

## 1150 Sectional Static Perimetry V<sub>tot</sub> (Hill of Vision)

| | | Sample Size (effective sample size after adjusting for inter-eye correlation $r=0.8$ ) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N=10 | | | | | | | | | |
| | (11) | (22) | (33) | (44) | (56) | (67) | (78) | (89) | (100) | (111) |
| SD=10 | 6.7 | 4.4 | 3.5 | 3.0 | 2.7 | 2.4 | 2.3 | 2.1 | 2.0 | 1.9 |
| SD=15 | 10.1 | 6.7 | 5.3 | 4.6 | 4.0 | 3.7 | 3.4 | 3.2 | 3.0 | 2.8 |
| SD=20 | 13.4 | 8.9 | 7.1 | 6.1 | 5.4 | 4.9 | 4.5 | 4.2 | 4.0 | 3.8 |
| SD=25 | 16.8 | 11.1 | 8.9 | 7.6 | 6.7 | 6.1 | 5.6 | 5.3 | 5.0 | 4.7 |

1151 Units = dB-sr

1152

1153

1154

1155

1156

1157

**Registry Sample Size Example** 

The following is an example of using the tables above and a set of assumptions for a given gene of interest to determine the precision of cross-sectional estimates of key measures.

| Gene | BBS1 | |
|---|---|---|
| Anticipated Sample Size | 50 | |
| Key Measure | Assumed Standard<br>Deviation (SD) | Precision around estimated mean value (half-width of 95% CI) |
| Visual Acuity | 10 | 2.7 |
| OCT EZ Area | 5 | 1.3 |
| SP Vtot | 20 | 5.4 |

1160 Assumptions based on Mean (standard deviation) of RUSH2A baseline V<sub>tot</sub>, VA, and OCT EZ RUSH2A shown below

| | Overall | USH2 | ARRP |
|---------------------|-------------|-------------|-------------|
| VA | 77.9 (11.7) | 76.5 (12.4) | 80.3 (10.2) |
| OCT EZ area | 3.6 (5.6) | 3.1 (5.7) | 4.3 (5.6) |
| SP V <sub>tot</sub> | 27.8 (23.7) | 22.5 (21.5) | 37.1 (24.7) |

#### 9.1.3 Natural History Study Sample Size Considerations

As noted in section 4.1, the designation of **NHS Target Genes** will be made by the Executive Committee on an ongoing basis and may depend on funding resources as well as Registry enrollment numbers within gene. The Natural History Study sample size for each gene will depend on the Registry enrollment. Since the within-gene Registry limit is 100 participants, this will be the maximum sample size for **NHS Target Genes**.

The following NHS sample size considerations focus on **NHS Objectives 1-3** (see section 1.3). For all of these objectives, the following principles will apply in the sections below:

- ➤ For simplicity across all measures, **percent change** will be considered for sample size justification purposes.
- Also for simplicity, although statistical analyses will include the data from each annual visit, **change from baseline to four (4) years** will be considered for sample size justification purposes.
- This simplistic approach will produce conservative estimates, in terms of precision. Future work will include exploring impact of sample sizes on these estimates when using all available longitudinal data, for example, how much will this improve precision. This will be documented separately.

1162

1163

1164

1165

1166

1167

1170

1171

1172

1173

1174

1175

1176

1177

#### NHS Objective 1 (Natural History)

- ➤ NHS Objective 1 is to characterize the natural history of retinal degeneration associated with disease-causing genetic variants over 4 years, using functional, structural, and patient-reported outcome measure, within gene.
- For a given gene, the potential sample size for the gene will impact the precision around the point estimates for changes in the outcome measures of interest.
- ➤ Table 9-5 provides the half-width of the 95% confidence interval (CI) around the estimated percent change in outcome measures under different possible sample sizes and standard deviations (SD) of the distribution of the percent change for any given outcome measure. The larger the SD and/or the smaller the sample size, the wider the CI, meaning the range of possible true values grows.

Table 9-5. Half-Width of 95% Confidence Intervals Around the Estimated Percent Change

| | | | (effective | e sample size | - | le Size ing for inter- | eve correlati | on r=0.8) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N=10 | N=20 | N=30 | N=40 | N=50 | N=60 | N=70 | N=80 | N=90 | N=100 |
| | (11) | (22) | (33) | (44) | (56) | (67) | (78) | (89) | (100) | (111) |
| SD=5% | 3% | 2% | 2% | 2% | 1% | 1% | 1% | 1% | 1% | 1% |
| SD=10% | 7% | 4% | 4% | 3% | 3% | 2% | 2% | 2% | 2% | 2% |
| SD=20% | 13% | 9% | 7% | 6% | 5% | 5% | 5% | 4% | 4% | 4% |
| SD=30% | 20% | 13% | 11% | 9% | 8% | 7% | 7% | 6% | 6% | 6% |
| SD=40% | 27% | 18% | 14% | 12% | 11% | 10% | 9% | 8% | 8% | 8% |
| SD=50% | 34% | 22% | 18% | 15% | 13% | 12% | 11% | 11% | 10% | 9% |
| SD=60% | 40% | 27% | 21% | 18% | 16% | 15% | 14% | 13% | 12% | 11% |

#### 

#### NHS Objective 2 (Structure-Function Relationship)

- ➤ NHS Objective 2 is to explore whether structural outcome measures can be validated as surrogates for functional outcomes in individuals with disease-causing genetic variants, within gene.
- For a given gene, the potential sample size for the gene will impact the precision around the point estimates for the correlation between the outcome measures of interest.
- ➤ Table 9-6 provides the 95% confidence intervals around the estimated correlation between outcome measures under different possible sample sizes and Pearson correlation coefficients.
  - O The Pearson correlation coefficient (r) can be used to assess the correlation between two different outcome measures. The distribution of r is not symmetric; therefore, CIs for the estimated correlation coefficient are not symmetric. A transformation of r (z = 0.5 \* ln ((1+r)/1-r)) is used to create a variable that is asymptotically distributed N (0, 1/(sqrt(N-3))) under the null hypothesis that r=0.

Table 9-6. 95% Confidence Intervals for an Observed Value of the Correlation between Outcome Measures.

| | | | (effectiv | ve sample size | _ | le Size | eye correlatio | n r = 0.8) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N=10 | N=20 | N=30 | N=40 | N=50 | N=60 | N=70 | N=80 | N=90 | N=100 |
| | (11) | (22) | (33) | (44) | (56) | (67) | (78) | (89) | (100) | (111) |
| r=0.3 | (-0.41,0.78) | (-0.16,0.66) | (-0.07,0.60) | (-0.01,0.56) | (0.02,0.53) | (0.05,0.51) | (0.07,0.50) | (0.09, 0.49) | (0.10,0.48) | (0.11,0.47) |
| r=0.4 | (-0.31,0.82) | (-0.05,0.72) | (0.05, 0.66) | (0.10,0.63) | (0.14,0.61) | (0.16,0.59) | (0.18,0.58) | (0.20,0.57) | (0.21, 0.56) | (0.22,0.55) |
| r=0.5 | (-0.19,0.86) | (0.07,0.77) | (0.17,0.73) | (0.22,0.70) | (0.26, 0.68) | (0.28, 0.67) | (0.30,0.66) | (0.31,0.65) | (0.33, 0.64) | (0.34,0.63) |
| r=0.6 | (-0.05,0.89) | (0.21,0.82) | (0.31,0.79) | (0.35,0.77) | (0.39,0.75) | (0.41,0.74) | (0.42,0.73) | (0.44,0.72) | (0.45, 0.72) | (0.46,0.71) |
| r=0.7 | (0.13,0.92) | (0.37,0.87) | (0.45,0.85) | (0.50,0.83) | (0.52,0.82) | (0.54,0.81) | (0.56,0.80) | (0.57,0.80) | (0.58, 0.79) | (0.58, 0.79) |
| r=0.8 | (0.34,0.95) | (0.55,0.92) | (0.62,0.90) | (0.65,0.89) | (0.67,0.88) | (0.69,0.88) | (0.70,0.87) | (0.70,0.87) | (0.71,0.86) | (0.72,0.86) |
| r=0.9 | (0.62,0.98) | (0.76,0.96) | (0.80,0.95) | (0.82,0.95) | (0.83,0.94) | (0.84,0.94) | (0.84,0.94) | (0.85,0.93) | (0.85,0.93) | (0.85,0.93) |

#### **NHS Objective 3 (Risk Factors for Progression)**

- NHS Objective 3 is to explore possible risk factors (genotype, phenotype, environmental, and comorbidities) for progression of the outcome measures at 4 years in individuals with disease-causing genetic variants, within gene.
- For a given gene, the potential sample size for the gene will impact the power to detect differences in changes from baseline among subgroups of interest.
- Figure 9-1 evaluates the <u>power to detect differences</u> in percent change from baseline to four (4) years among two (2) subgroups of equally distributed sizes, under various assumptions of true mean difference (x-axis) and standard deviation (SD) of the distribution of percent change. If subgroups are not equally sized, the smallest detectable difference (with the same power) will be larger. All calculations are based on a Type I ( $\alpha$ ) error rate of 0.05.
  - o For example, with a total sample size of twenty (20), assuming ten (10) in each of two (2) subgroups, to have power of 80% or more, the true difference needs to be approximately 1.25 SDs (a mean difference of 25% if the SD of the percent change over four (4) years 20%)
- ➤ **Also Note:** <u>Within-subgroup</u> point estimates and CIs will also be important. **Table 9-3** above can be applied to potential subgroup sample sizes as well to consider the precision that would be observed.

#### Figure 9-1 Power to Detect Differences in Subgroups



1234



#### NHS Sample Size Example

1236

1237

1238

The following is an example template of using the tables above and a set of assumptions for a given gene of interest to determine the impact on NHS Objectives.

| Target Gene | MYO7A |
|---|---|
| Target Sample Size | 50 |
| Data to consider for | <u>Data</u> |
| assumptions | • RUSH2A Data – Mean (SD) percent change at 24M |
| | <ul> <li>Visual Acuity: -2.3 (5.1)%</li> </ul> |
| | o OCT EZ area: -2.2 (21.8)% |
| | o Static Perimetry HOV: -12.4 (28.2)% |
| | Assume: |
| | • Inter-eye correlation = 0.8 |
| | <ul> <li>SD for percent change at 4 years</li> </ul> |
| | ○ Visual Acuity → 5% |
| | $\circ$ OCT EZ area $\rightarrow$ 20% |
| | <ul> <li>Static Perimetry HOV → 30%</li> </ul> |
| | · |

| NHS Objective 1 (Natural | The half-width of a 95% CI around the point estimate for mean | | |
|---|---|---|---|
| History) | percent change at 4 years would be | | |
| | Visual Acuity | Visual Acuity OCT EZ area Static Pe | |
| | 1% | 5% | 8% |
| NHS Objective 2 (Structure- | The 95% CI around co | rrelation between an | ny two outcome measures |
| Function Relationship) | would be | | |
| | if the observed corre | elation r = 0.3 | (0.02, 0.53) |
| | if the observed correlation $r = 0.5$ (0.26, 0.68) | | |
| | if the observed correlation $r = 0.8$ (0.67, 0.88) | | |
| NHS Objective 3 (Risk | A comparison of two e | | |
| <b>Factors for Progression)</b> | | power to conclude | there is a difference if the |
| | true difference is | | |
| | Visual Acuity OCT EZ area Static Perimetry HOV | | |
| | 4% 15% 23%* | | |
| | [Type I ( $\alpha$ ) error rate of 0.05] | | |
| | * For example, if one subgroup had a percent change of 13%, the | | |
| | other subgroup would need a percent change of 36% to statistically | | |
| | conclude there is a diff | erence. | |

#### 1239

1240

1244

1245

1246

1247

#### 9.2 Data Analysis

- The analysis plans below are written with respect to the majority of outcomes of interest.
- Analyses will include data on both eyes for each participant, and confidence intervals will adjust for correlation between two (2) eyes of the same participant.

#### 9.2.1 Registry Data Analysis

The following Registry data analysis considerations focus on **Registry Objective 2** (see section 1.3). Applicability of <u>within-gene</u> objectives will depend on <u>within-gene</u> sample size as noted below. <u>If less than 20</u>, limit primary objective to describing the cohort in the form of case histories. Objectives may still be explored depending on the needs for a specific gene.

12481249

1250

1251

1252

1253

1254

1255

1256

1257

### Registry Objective 2 (Cross-Sectional Phenotype Characterization)

- Registry Objective 2 is to characterize cross-sectional retinal dystrophy associated with disease-causing genetic variants using functional and structural measures (visual acuity, OCT, static perimetry), within-gene. Structure-function relationships and risk factors for disease severity will also be explored within-gene.
  - The distribution of each cross-sectional outcome measure will be summarized (including tabulating categorically, as well as means, SDs, medians, quartiles, ranges; where sample size 20 or more).

| 1258<br>1259 | | Scatterplots and Spearman correlation coefficients between cross-sectional outcome measures will be explored ( <i>where sample size is 20 or more</i> ) |
|---|---|---|
| 1260<br>1261<br>1262 | f | Possible risk factors (genotype, phenotype, environmental, and comorbidities) For cross-sectional outcome measures will be explored ( <i>where sample size is 40 or more</i> ). |
| 1263<br>1264<br>1265<br>1266<br>1267<br>1268<br>1269 | | Methods will include univariate and multivariate analysis of<br>covariance (ANCOVA) models. A stepwise selection procedure will<br>be used to build the final model. A threshold of P<0.10 will be used to<br>add to the model, and a threshold of P<0.05 will be used to remain in<br>the multivariate model. Linearity of continuous factors will be<br>assessed, and possibly quadratic or cubic terms will be considered if<br>non-linear. |
| 1270 | | <ul> <li>Potential risk factors to evaluate include:</li> </ul> |
| 1271 | | Phenotypic: |
| 1272<br>1273<br>1274<br>1275<br>1276 | | <ul> <li>Clinical diagnosis (if applicable)</li> <li>Duration of disease</li> <li>Age of onset of initial vision symptoms</li> <li>Gender</li> <li>Race/ethnicity</li> </ul> |
| 1277 | | Visual acuity |
| 1278 | | <ul> <li>Lens Status (phakic/pseudophakic/aphakic)</li> </ul> |
| 1279 | | ■ Genotypic: |
| 1280 | | <ul> <li>Characterizations of the variants</li> </ul> |
| 1281 | | <ul><li>Environmental factors</li></ul> |
| 1282<br>1283<br>1284<br>1285 | | <ul> <li>Smoking status</li> <li>Vitamin A use</li> <li>Docosahexaenoic acid (DHA) use</li> <li>Lutein use</li> </ul> |
| 1286<br>1287<br>1288<br>1289<br>1290<br>1291<br>1292<br>1293 | r<br>e<br>r<br>r<br>v | Variability of symmetry of left and right eye cross-sectional outcome measures will be evaluated by scatterplots. Bland-Altman plots of the intereye difference versus the mean value will be inspected and a linear regression model for the differences will be used to test whether the intercept (overall mean difference) and slope is 0. The plot will be inspected to evaluate whether variability between eyes changes with greater mean values. The intraclass correlation coefficient of the values and the within-person variance will be estimated. |
| 1294 | 9.2.2 Natural H | History Data Analysis |
| 1295 | The following Natu | aral History Study data analysis considerations focus on NHS Objectives 1-3 |
| 1296 | | pplicability of within-gene objectives will depend on within-gene sample size |

as noted below. <u>If less than 20,</u> limit primary objective to describing the cohort in the form of case histories. Objectives may still be explored depending on the needs for a specific gene.

#### **NHS Objective 1 (Natural History)**

- ➤ NHS Objective 1 is to characterize the natural history of retinal degeneration associated with disease-causing genetic variants over 4 years, using functional, structural, and patient-reported outcome measure, <u>within-gene</u> (where sample size 20 or more).
  - O Analysis plan for functional and structural measures: The distribution of each outcome at each visit will be summarized (including tabulating categorically, as well as means, SDs, medians, quartiles, ranges; both the absolute change and percent change will be evaluated, tests performed multiple times will be analyzed using average of all available tests). To determine the average annual rate of progression in the population for each outcome, a repeated measure least squares regression model will be fit using all available outcome data at baseline and all annual visits. Multiple imputation will be used to impute the outcome values for all missing time points (including participants who discontinue follow up prior to 48 months). Secondary analyses using binary definitions of outcome measures will also be explored in time to event analyses; Kaplan-Meier estimates with 95% confidence intervals will be calculated.
  - O Analysis plan for PRO measures: The scoring of each questionnaire will be completed according to the procedures for each instrument and is detailed further in a separate statistical analysis plan. Baseline scores will be cross tabulated with categorical (severity of disease) versions of the outcome measures of interest at baseline. Changes in scores will be cross tabulated with binary (progression of disease) versions of the outcome measures of interest at the 24- and 48-month visits. A generalized linear model adjusted for baseline differences will be explored.

#### NHS Objective 2 (Structure-Function Relationship)

- > NHS Objective 2 is to explore whether structural outcome measures can be validated as surrogates for functional outcomes in individuals with disease-causing genetic variants, within gene (where sample size 20 or more).
  - Analysis plan: Scatterplots and Spearman correlation coefficients of changes in functional and structural outcome measures of progression from baseline to each visit will be evaluated.

#### **NHS Objective 3 (Risk Factors for Progression)**

- ➤ NHS Objective 3 is to explore possible risk factors (genotype, phenotype, environmental, and comorbidities) for progression of the outcome measures at 4 years in individuals with disease-causing genetic variants, within-gene (where sample size 40 or more).
  - Analysis plan: The distribution of each outcome in terms of both absolute change and percent change from baseline to 4 years will be summarized (including tabulating categorically, as well as means, standard deviations,

| 1339<br>1340 | medians, quartiles), stratified by categorical levels of each potential risk factor of interest (listed below). Potential risk factors to evaluate include: |
|---|---|
| 1341 | o Phenotypic: |
| 1342<br>1343<br>1344<br>1345<br>1346<br>1347<br>1348 | <ul> <li>Clinical diagnosis (if applicable)</li> <li>Duration of disease</li> <li>Age of onset of initial vision symptoms</li> <li>Gender</li> <li>Race/ethnicity</li> <li>Visual Acuity</li> <li>Lens Status (phakic/pseudophakic/aphakic)</li> </ul> |
| 1349 | o Genotypic: |
| 1350 | <ul> <li>Characterizations of the variants</li> </ul> |
| 1351 | <ul> <li>Environmental factors</li> </ul> |
| 1352<br>1353<br>1354<br>1355 | <ul> <li>Smoking status at baseline</li> <li>Vitamin A use at baseline</li> <li>Docosahexaenoic acid (DHA) use at baseline</li> <li>Lutein use at baseline</li> </ul> |
| 1356 | Other Planned Analyses |
| 1357<br>1358<br>1359<br>1360<br>1361<br>1362<br>1363<br>1364<br>1365<br>1366<br>1367 | <ul> <li>Analysis plan for variability of repeat perimetry testing at baseline: Scatterplots and Spearman correlation coefficients for pairs (first versus second) of testing values for each repeated perimetry test. Bland-Altman plots of difference versus the mean value will be inspected. The intraclass correlation coefficient of the values and the within-eye variance will be estimated.</li> <li>Analysis plan for the symmetry of left eye versus right eye: At baseline and each subsequent testing time, the symmetry of the test result values from the left and right eyes will be assessed and the symmetry of the change from baseline from the left and right eyes will be assessed for each follow-up visit. Bland-Altman plots of the inter-eye difference versus the mean value will be inspected. The intraclass correlation coefficient of the values will be estimated.</li> </ul> |
| 1368 <b>9.2</b> | .3 Interim Data Analysis |
| 1369<br>1370<br>1371 | No formal interim analysis or "stopping guidelines" are planned for determining early stopping according to statistical rules, as no intervention is being studied and thus early efficacy and safety signals are not applicable. |
| 1372<br>1373<br>1374<br>1375 | Interim analyses will be planned for other reasons, including to evaluate data at baseline and annual visits for reporting in preliminary manuscripts, as well as monitoring data for recruitment and retention benchmarks, and quality assurance throughout the duration of the study. The FFB Consortium Executive Committee will review and oversee these data and their use in reporting. |

| 1377 | <b>Chapter 10: Data Collection and Monitoring</b> |
|---|---|
| 1378 | 10.1 Case Report Forms and Other Data Collection |
| 1379<br>1380<br>1381<br>1382<br>1383<br>1384<br>1385<br>1386 | The main study data are collected on electronic case report forms (eCRFs). When data are directly collected in electronic case report forms, this will be considered the source data. For any data points for which the eCRF is not considered source (e.g., lab results that are transcribed from a printed report into the eCRF), the original source documentation must be maintained in the participant's study chart or medical record. <b>This source must be readily verifiable against the values entered into eCRF.</b> Even where all study data are directly entered into the eCRFs at office visits, evidence of interaction with a live subject must be recorded (e.g., office note, visit record, etc.) and provided to the coordinating center for review. |
| 1387<br>1388<br>1389<br>1390 | Each participating site will maintain appropriate medical and research records for this trial, in compliance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) E6 and regulatory and institutional requirements for the protection of confidentiality of participants |
| 1391 | 10.1.1 Central Genetics Auditor (CGA) |
| 1392<br>1393<br>1394 | The CGA will review the genetic lab report(s) submitted by the clinical site during genetic screening and will document their verification of these genetic data on the FFB Consortium study website. |
| 1395 | 10.1.2 Genetics Committee (GC) |
| 1396<br>1397<br>1398<br>1399 | In addition to providing assistance in the interpretation/evaluation of whether the mutations are causative of the disease on the FFB Consortium study website, the Genetics Committee will review and provide approval for the use of genetic reports from research labs to be used for determining participant eligibility. |
| 1400 | 10.1.3 Reading Center (RC) |
| 1401<br>1402<br>1403<br>1404 | Reading Centers will conduct grading of the study data collected using the FFB Consortium study website. The Reading Centers will provide the graded data through a data transfer or by entering the graded data on the study website. These data will remain in the study database and will not be provided to the clinical site. |
| 1405 | 10.2 Study Records Retention |
| 1406<br>1407<br>1408 | Each participating site will maintain appropriate medical and research records for this trial, in compliance with ICH E6 and regulatory and institutional requirements for the protection of confidentiality of participants. |
| 1409<br>1410<br>1411<br>1412<br>1413 | Study documents will be retained for a minimum of six (6) years from the date on which the CC receives IRB approval to close the study. These documents should be retained for a longer period, however, if required by local regulations. No records will be destroyed without the written consent of the Sponsor. It is the responsibility of the Sponsor to inform the Principal Investigator (PI) when these documents no longer need to be retained. |

#### 10.3 Quality Assurance and Monitoring

- Designated personnel from the Coordinating Center will be responsible for maintaining quality
- assurance (QA) and quality control (QC) systems to ensure that the clinical portion of the trial is
- 1417 conducted and data are generated, documented and reported in compliance with the protocol,
- Good Clinical Practice (GCP) and the applicable regulatory requirements, as well as to ensure
- that the rights and wellbeing of trial participants are protected and that the reported trial data are
- accurate, complete, and verifiable.

1414

1431

1432

1433

1434

1435

1436

1438

1440

1449

- 1421 A risk-based monitoring (RBM) plan will be developed and revised as needed during the study,
- consistent with the FDA "Guidance for Industry Oversight of Clinical Investigations A Risk-
- Based Approach to Monitoring" (August 2013). Study conduct and monitoring will conform
- with 21 Code of Federal Regulations (CFR) 312.<sup>10</sup> This plan describes in detail who will conduct
- the monitoring, at what frequency monitoring will be done, at what level of detail monitoring
- will be performed, and the distribution of monitoring reports.
- The data of most importance for monitoring at the site are participant eligibility and adverse
- events. Therefore, the RBM plan will focus on these areas. As much as possible, remote
- monitoring will be performed in real-time with on-site monitoring performed to evaluate the
- verity and completeness of the key site data. Elements of the RBM may include:
  - Qualification assessment, training, and certification for sites and site personnel
    - Oversight of Institutional Review Board (IRB) coverage and informed consent procedures
      - Central (remote) data monitoring: validation of data entry, data edits/audit trail, protocol review of entered data and edits, statistical monitoring, study closeout
      - On-site monitoring (site visits): source data verification, site visit report
- ◆ Communications with site staff
  - Patient retention and visit completion
- Quality control reports
  - Management of noncompliance
- ◆ Documenting monitoring activities
- ◆ Adverse event reporting and monitoring
- 1443 Coordinating Center representatives or their designees may visit the study facilities at any time in
- order to maintain current and personal knowledge of the study through review of records,
- 1445 comparison with source documents, observation and discussion of the conduct and progress of
- the study. The investigational site will provide direct access to all trial-related sites, source
- data/documents, and reports for the purpose of monitoring and auditing by the Sponsor, and
- inspection by local and regulatory authorities.

#### 10.4 Protocol Deviations

- A protocol deviation is any noncompliance with the clinical trial protocol, GCP, or procedure
- requirements. The noncompliance may be either on the part of the participant, the Investigator(s),
- or the study site staff.

| 1453 | A significant (or major) deviation is any deviation that departs from the established materials in |
|---|---|
| 1454 | such a way that it poses an increase in the risk to the study participants, adversely affects the |
| 1455 | welfare, rights, or safety of the research study participants, or negatively influences the scientific |
| 1456<br>1457 | study integrity. As a result of significant deviations, corrective and preventive actions are to be developed by the site and implemented promptly. |
| 1458<br>1459 | The site Principal Investigator (PI) and study staff are responsible for knowing and adhering to their IRB/EC requirements. |

#### **Chapter 11: Ethics/Protection of Human Participants** 1460 11.1 Ethical Standard 1461 The Principal Investigator (PI) will ensure that this study is conducted in full conformity with 1462 1463 Regulations for the Protection of Human Participants of Research in accordance with ICF E6/GCP, EC requirements, and local laws and regulations, as applicable. 1464 1465 11.2 Institutional Review Boards 1466 The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the IRB for review and approval. Approval of both the protocol and the consent 1467 1468 form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. All 1469 changes to the consent form will be IRB approved; a determination will be made regarding 1470 whether previously consented participants need to be re-consented. 1471 11.3 Informed Consent Process 1472 11.3.1 Consent Procedures and Documentation 1473 Informed consent is a process that is initiated prior to the individual's agreeing to participate in 1474 1475 the study and continues throughout the individual's study participation. Extensive discussion of risks and possible benefits of participation will be provided to the participants and their families. 1476 Consent forms will be IRB/EC-approved, and the participant will be asked to read and review the 1477 document. The Investigator(s) will explain the research study to the participant and answer any 1478 questions that may arise. All participants will receive a verbal explanation in terms suited to their 1479 comprehension of the purposes, procedures, and potential risks of the study and of their rights as 1480 research participants. Participants will have the opportunity to carefully review the written 1481 consent form and ask questions prior to signing. 1482 1483 The participants will have the opportunity to discuss the study with their surrogates or think about it prior to agreeing to participate. The participant will sign the informed consent document 1484 prior to any procedures being done specifically for the study. The participants may withdraw 1485 consent at any time throughout the course of the trial. A copy of the informed consent document 1486 will be given to the participants for their records. The rights and welfare of the participants will 1487 be protected by emphasizing to them that the quality of their medical care will not be adversely 1488 1489 affected if they decline to participate in this study. 11.3.2 Participant and Data Confidentiality 1490 Participant confidentiality is strictly held in trust by the participating Investigator(s), their staff, 1491 1492 and the Sponsor(s) and their agents. This confidentiality is extended to cover use of genetic tests in addition to the clinical information relating to participants. Therefore, the study protocol, 1493 1494 documentation, data, and all other information generated will be held in strict confidence. No 1495 information concerning the study, or the data will be released to any unauthorized third party without prior written approval of the Sponsor. 1496

The study monitor, other authorized representatives of the Sponsor, representatives of the IRB/EC, regulatory agencies or company supplying study product may inspect all documents

1497

and records required to be maintained by the Principal Investigator, including but not limited to, 1499 1500 medical records (office, clinic, or hospital) for the participants in this study. The clinical study site will permit access to such records. 1501 The study participant's contact information will be securely stored at each clinical site for 1502 internal use during the study. At the end of the study, all records will continue to be kept in a 1503 1504 secure location for as long a period as dictated by the reviewing IRB/EC, institutional policies, or Sponsor requirements. 1505 1506 Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the FFB Consortium Coordinating Center, located 1507 at the Jaeb Center for Health Research in Tampa, FL. This will not include the participant's 1508 contact or identifying information, unless otherwise specified in the informed consent form. 1509 Rather, individual participants and their research data will be identified by a unique study 1510 identification number. The study data entry and study management systems used by clinical sites 1511 and by the FFB Consortium Coordinating Center research staff will be secured and password 1512 protected. At the end of the study, all study databases will be de-identified and archived at the 1513 FFB Consortium Coordinating Center. 1514 11.3.3 Future Use of Data and Ocular Images 1515 Data and images collected for this study will be analyzed and stored at the FFB Coordinating 1516 Center and the Reading Centers. After the study is completed, the de-identified, archived data 1517 will be transmitted to and stored at the FFB Consortium Coordinating Center, under the 1518 supervision of the Protocol Director, for use by other researchers including those outside of the 1519

study. Permission to transmit data to the FFB Consortium Coordinating Center will be included

1520

1521

in the informed consent.

| 1522 | | Chapter 12: References |
|---|---|---|
| 1523 | | References |
| 1524 | | |
| 1525 | 1. | Sahel JA, Bennett J, Roska B. Depicting brighter possibilities for treating blindness. Sci |
| 1526 | | <i>Transl Med.</i> 2019;11(494). |
| 1527 | 2. | Scholl HP, Strauss RW, Singh MS, et al. Emerging therapies for inherited retinal |
| 1528 | | degeneration. Sci Transl Med. 2016;8(368):368rv366. |
| 1529 | 3. | Duncan JL, Pierce EA, Laster AM, et al. Inherited Retinal Degenerations: Current |
| 1530 | | Landscape and Knowledge Gaps. Transl Vis Sci Technol. 2018;7(4):6. |
| 1531 | 4. | Thompson DA, Iannaccone A, Ali RR, et al. Advancing Clinical Trials for Inherited |
| 1532 | | Retinal Diseases: Recommendations from the Second Monaciano Symposium. Transl Vis |
| 1533 | | Sci Technol. 2020;9(7):2. |
| 1534 | 5. | Csaky K, Ferris F, 3rd, Chew EY, Nair P, Cheetham JK, Duncan JL. Report From the |
| 1535 | | NEI/FDA Endpoints Workshop on Age-Related Macular Degeneration and Inherited |
| 1536 | | Retinal Diseases. Invest Ophthalmol Vis Sci. 2017;58(9):3456-3463. |
| 1537 | 6. | Sahel JA, Grieve K, Pagot C, et al. Assessing Photoreceptor Status in Retinal |
| 1538 | | Dystrophies: From High-Resolution Imaging to Functional Vision. Am J Ophthalmol. |
| 1539 | | 2021;230:12-47. |
| 1540 | 7. | Cideciyan AV, Krishnan AK, Roman AJ, Sumaroka A, Swider M, Jacobson SG. |
| 1541 | | Measures of Function and Structure to Determine Phenotypic Features, Natural History, |
| 1542 | | and Treatment Outcomes in Inherited Retinal Diseases. Annu Rev Vis Sci. 2021;7:747- |
| 1543 | | 772. |
| 1544 | 8. | Food and Drug Administration. Rare Diseases: Natural History Studies for Drug |
| 1545 | | Development. In. Draft Guidance for Industry, 2019. |
| 1546 | 9. | Food and Drug Administration. Guidance for Industry Oversight of Clinical |
| 1547 | | Investigations - A Risk-Based Approach to Monitoring. In:2013. |
| 1548 | 10. | Food and Drug Administration. 21 Code of Federal Regulations (CFR) 312. In:2022. |
| 1549 | | |